CLINICAL TRIAL: NCT05415215
Title: A Phase IIIB, Multinational, Multicenter, Randomized, Open-Label Study to Evaluate Patient Preference for Home Administration of Fixed-Dose Combination of Pertuzumab and Trastuzumab for Subcutaneous Administration in Participants With Early or Locally Advanced/Inflammatory HER2-Positive Breast Cancer
Brief Title: A Study to Evaluate Patient Preference for Home Administration of Fixed-Dose Combination of Pertuzumab and Trastuzumab for Subcutaneous Administration in Participants With Early or Locally Advanced/Inflammatory HER2-Positive Breast Cancer
Acronym: ProHer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MO43110; 2021-002346-33 (EudraCT Number); 2023-506380-33-00 (EU CTIS Number)
Record Dates: First submitted 2022-06-08; First posted 2022-06-13 (Actual); Results first posted 2026-01-12 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Early Breast Cancer; Locally Advanced Breast Cancer; Inflammatory Breast Cancer
Keywords: patient preference; home administration; fixed-dose combination of pertuzumab and trastuzumab; subcutaneous administration
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms; Patient Preference | interventions — Trastuzumab; Injections, Subcutaneous; pertuzumab; Ado-Trastuzumab Emtansine; Surgical Procedures, Operative; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Arm A: Pertuzumab IV and Trastuzumab IV Plus Investigator's Choice of Chemotherapy (Other): During the neoadjuvant phase, the enrolled participants randomized to this arm will receive treatment with pertuzumab and trastuzumab intravenously (PH IV) plus investigator's choice of chemotherapy (Option 1, 2, or 3). With chemotherapy Option 1, PH IV will be administered at each cycle from Cycles 1 to 6 (1 cycle is 3 weeks); with chemotherapy Options 2 and 3, PH IV will be administered once per cycle from Cycles 5 to 8 (1 cycle is 3 weeks).
  Interventions: Drug: Pertuzumab IV; Drug: Trastuzumab IV; Drug: Investigator's Choice of Chemotherapy; Procedure: Surgery; Radiation: Radiotherapy
- Arm B: PH FDC SC Plus Investigator's Choice of Chemotherapy (Other): During the neoadjuvant phase, the enrolled participants randomized to this arm will receive treatment with the fixed dose combination of pertuzumab and trastuzumab for subcutaneous use (PH FDC SC) plus investigator's choice of chemotherapy (Option 1, 2, or 3). With chemotherapy Option 1, PH FDC SC will be administered at each cycle from Cycles 1 to 6 (1 cycle is 3 weeks); with chemotherapy Options 2 and 3, PH FDC SC will be administered once per cycle from Cycles 5 to 8 (1 cycle is 3 weeks).
  Interventions: Drug: Fixed Dose Combination of Pertuzumab and Trastuzumab for Subcutaneous Use (PH FDC SC); Drug: Investigator's Choice of Chemotherapy; Procedure: Surgery; Radiation: Radiotherapy
- Arm C: Adjuvant PH FDC SC in Hospital, Then at Home (Experimental): During the adjuvant phase, participants who have achieved pCR after surgery will be treated with 2 cycles of PH FDC SC in the hospital (run-in period). After completion of the last cycle of radiotherapy and the last cycle of PH FDC SC (run-in period), participants will then be randomized with a ratio of 1:1 into one of two treatment arms (Arm C or D) in a cross-over treatment period to receive the next 6 cycles of PH FDC SC treatment. Participants in Arm C will receive 3 cycles of PH FDC SC in the hospital and then 3 cycles of PH FDC SC in the home setting. After the cross-over treatment period, participants will receive the remaining PH FDC SC treatment cycles required to complete the planned 18 cycles of HER2-directed therapy, unless of disease recurrence, unacceptable toxicity, or withdrawal. Study treatment during this treatment continuation period will be administered either in the hospital or in the home setting as selected by the participant at the end of the crossover period.
  Interventions: Drug: Fixed Dose Combination of Pertuzumab and Trastuzumab for Subcutaneous Use (PH FDC SC)
- Arm D: Adjuvant PH FDC SC at Home, Then in Hospital (Experimental): During the adjuvant phase, participants who have achieved pCR after surgery will be treated with 2 cycles of PH FDC SC in the hospital (run-in period). After completion of the last cycle of radiotherapy and the last cycle of PH FDC SC (run-in period), participants will then be randomized with a ratio of 1:1 into one of two treatment arms (Arm C or D) in a cross-over treatment period to receive the next 6 cycles of PH FDC SC treatment. Participants in Arm D will receive 3 cycles of PH FDC SC in the home setting and then 3 cycles of PH FDC SC in the hospital. After the cross-over treatment period, participants will receive the remaining PH FDC SC treatment cycles required to complete the planned 18 cycles of HER2-directed therapy, unless of disease recurrence, unacceptable toxicity, or withdrawal. Study treatment during this treatment continuation period will be administered either in the hospital or in the home setting as selected by the participant at the end of the crossover period.
  Interventions: Drug: Fixed Dose Combination of Pertuzumab and Trastuzumab for Subcutaneous Use (PH FDC SC)
- Arm E: Adjuvant Trastuzumab Emtansine (Other): Participants with pathological evidence of residual invasive carcinoma in the breast or axillary lymph nodes following completion of preoperative therapy and surgery will enter Arm E to receive trastuzumab emtansine for 14 cycles. Trastuzumab emtansine will be administered IV in the hospital as per prescribing information.
  Interventions: Drug: Trastuzumab Emtansine

INTERVENTIONS:
Drug: Fixed Dose Combination of Pertuzumab and Trastuzumab for Subcutaneous Use (PH FDC SC) — PH FDC SC is administered subcutaneously (SC) as a fixed non-weight-based dose. A loading dose of 1200 milligram (mg) pertuzumab, 600 mg trastuzumab, and 30,000 units of recombinant human PH20 hyaluronidase (rHuPH20) is given in the first cycle (1 cycle is 21 days). In subsequent cycles, maintenance doses of 600 mg pertuzumab, 600 mg trastuzumab, and 20,000 units rHuPH20 are administered once every 3 weeks (Q3W).
  Other Names: PHESGO®; Pertuzumab, Trastuzumab, and Hyaluronidase-zzxf; Pertuzumab, Trastuzumab, and rHuPH20; RO7198574; RG6264
  Arms: Arm B: PH FDC SC Plus Investigator's Choice of Chemotherapy; Arm C: Adjuvant PH FDC SC in Hospital, Then at Home; Arm D: Adjuvant PH FDC SC at Home, Then in Hospital
Drug: Pertuzumab IV — Pertuzumab is given as a fixed dose of 840 mg intravenous (IV) loading dose and then 420 mg IV for subsequent maintenance doses once every 3 weeks.
  Other Names: Perjeta®; RO4368451
  Arms: Arm A: Pertuzumab IV and Trastuzumab IV Plus Investigator's Choice of Chemotherapy
Drug: Trastuzumab IV — Trastuzumab is given as an 8 milligram per kilogram (mg/kg) intravenous (IV) loading dose and then 6 mg/kg IV for subsequent maintenance doses once every 3 weeks.
  Other Names: Herceptin®; RO0452317
  Arms: Arm A: Pertuzumab IV and Trastuzumab IV Plus Investigator's Choice of Chemotherapy
Drug: Trastuzumab Emtansine — Trastuzumab emtansine will be given at a dose of 3.6 mg/kg by intravenous (IV) infusion, once every 3 weeks.
  Other Names: Kadcyla®; ado-trastuzumab emtansine; T-DM1; RO5304020
  Arms: Arm E: Adjuvant Trastuzumab Emtansine
Drug: Investigator's Choice of Chemotherapy — Option 1: Docetaxel and carboplatin once every 3 weeks for 6 cycles; Option 2: Doxorubicin plus cyclophosphamide once every 3 weeks for 4 cycles, followed by a taxane (docetaxel once every 3 weeks for 4 cycles or paclitaxel once every week for 12 cycles); Option 3: Dose-dense doxorubicin plus cyclophosphamide (ddAC) once every 2 weeks for 4 cycles, followed by a taxane (docetaxel once every 3 weeks for 4 cycles or paclitaxel once every week for 12 cycles).
  Arms: Arm A: Pertuzumab IV and Trastuzumab IV Plus Investigator's Choice of Chemotherapy; Arm B: PH FDC SC Plus Investigator's Choice of Chemotherapy
Procedure: Surgery — After completing their neoadjuvant therapy, participants will undergo surgical resection for early or locally advanced HER2+ breast cancer (if eligible for surgery). Participants may undergo breast-conserving surgery or mastectomy according to routine clinical practice. The surgery cannot be performed ≤2 weeks from the last systemic neoadjuvant therapy and must be performed ≤6 weeks after the last systemic neoadjuvant therapy.
  Arms: Arm A: Pertuzumab IV and Trastuzumab IV Plus Investigator's Choice of Chemotherapy; Arm B: PH FDC SC Plus Investigator's Choice of Chemotherapy
Radiation: Radiotherapy — After surgery, radiotherapy is to be given as clinically indicated and as per local practice or institutional standards. The selected radiotherapy regimen should be initiated within 4 weeks after surgery.
  Arms: Arm A: Pertuzumab IV and Trastuzumab IV Plus Investigator's Choice of Chemotherapy; Arm B: PH FDC SC Plus Investigator's Choice of Chemotherapy

SUMMARY:
This is a Phase IIIb, multinational, multicenter, randomized, open-label study to evaluate patient preference of the fixed-dose combination of pertuzumab and trastuzumab for subcutaneous use (PH FDC SC) administration in the home setting compared with the hospital setting during the cross-over period of adjuvant treatment in participants with early or locally advanced/inflammatory human epidermal growth factor receptor 2-positive (HER2+) breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Intact skin at planned site of subcutaneous (SC) injections
* Left ventricular ejection fraction (LVEF) greater than or equal to (≥)55% by echocardiogram (ECHO) or multiple-gated acquisition scan (MUGA)
* Negative human immunodeficiency virus (HIV) test at screening
* Negative hepatitis B surface antigen (HBsAg) test at screening
* Positive hepatitis B surface antibody (HBsAb) test at screening, or negative HBsAb at screening accompanied by either of the following: Negative total hepatitis B core antibody (HBcAb); Positive total HBcAb test followed by a negative (per local laboratory definition) hepatitis B virus (HBV) DNA test
* Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening
* For female participants of childbearing potential: agreement to remain abstinent or use contraception and agree to refrain from donating eggs during the treatment period and for 7 months after the final dose of the study treatment
* For male participants: agreement to remain abstinent or use a condom, and agree to refrain from donating sperm during the treatment period and for 7 months after the final dose of study treatment

Disease-specific Inclusion Criteria:

* Female and male participants with stage II-IIIC early or locally advanced/inflammatory human epidermal growth factor receptor 2-positive (HER2+) breast cancer
* Primary tumor >2 centimetres (cm) in diameter, or node-positive disease
* HER2+ breast cancer confirmed by a local laboratory prior to study enrollment. HER2+ status will be determined based on pretreatment breast biopsy material and defined as 3+ by Immunohistochemistry (IHC) and/or positive by HER2 amplification by in situ hybridization (ISH) following American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines 2018 and updates (Wolff et al. Arch Pathol Lab Med 2018)
* Hormone receptor status of the primary tumor determined by local assessment following American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines and updates (Allison et al. J Clin Oncol 2020)
* Agreement to undergo mastectomy or breast conserving surgery after neoadjuvant therapy, including the axillary nodes
* Availability of formalin-fixed, paraffin-embedded (FFPE) tumor tissue block for local confirmation of HER2 and hormone receptor status following current ASCO/CAP guidelines

Inclusion Criteria for Treatment with Adjuvant PH FDC SC:

* Completed the neoadjuvant phase of this study and underwent surgery, and achieved pathologic complete response (pCR), defined as eradication of invasive disease in the breast and axilla according to the current American Joint Committee on Cancer (AJCC) staging system classification, and using the resected specimen by the local pathologist on the basis of guidelines to be provided in a pathology manual
* Adequate wound healing after breast cancer surgery per investigator's assessment to allow initiation of study treatment within less than or equal to (≤)9 weeks of last systemic neoadjuvant therapy

Exclusion Criteria:

* Stage IV (metastatic) breast cancer
* History of concurrent or previously treated non-breast malignancies, except for appropriately treated 1) non-melanoma skin cancer and/or 2) in situ carcinomas, including cervix, colon, and skin. A participant with previous invasive non-breast cancer is eligible provided he/she has been disease free for more than 5 years
* Participants who are pregnant or breastfeeding or intending to become pregnant during the study or within 7 months after the final dose of study treatments
* Treatment with investigational therapy within 28 days prior to initiation of study treatment
* Active, unresolved infections at screening requiring treatment
* Participants who may have had a recent episode of thromboembolism and are still trying to optimize the anticoagulation dose and/or have not normalized their International Normalized Ratio (INR)
* Serious cardiac illness or medical conditions
* History of ventricular dysrhythmias or risk factors for ventricular dysrhythmias
* Inadequate bone marrow function
* Impaired liver function
* Renal function with creatinine clearance <50 mL/min using the Cockroft-Gault formula and serum creatinine >1.5x upper limit of normal (ULN)
* Major surgical procedure unrelated to breast cancer within 28 days prior to study entry or anticipation of the need for major surgery during the course of study treatment
* Current severe, uncontrolled systemic disease that may interfere with planned treatment
* Any serious medical condition or abnormality in clinical laboratory tests that precludes an individual's safe participation in and completion of the study
* Treatment with a live vaccine (e.g., FluMist) in the 30 days prior to initiation of study treatment, or anticipation of need for such a vaccine during treatment or within 90 days after the final dose of study treatment
* Known active liver disease, for example, active viral hepatitis infection, autoimmune hepatic disorders, or sclerosing cholangitis
* Known hypersensitivity to any of the study drugs, excipients, and/or murine proteins or a history of severe allergic or immunological reactions, e.g., difficult to control asthma
* Current chronic daily treatment with corticosteroids
* Assessment by the investigator as being unable or unwilling to comply with the requirements of the protocol

Cancer-specific Exclusion Criteria for Neoadjuvant Phase:

* Participants who have received any previous systemic therapy for treatment or prevention of breast cancer, or previous chest irradiation for the treatment of cancer
* Participants who have a past history of ductal carcinoma in situ (DCIS) or lobular carcinoma in situ (LCIS) if they have received any systemic therapy for its treatment or radiation therapy to the ipsi- or contralateral breast cancer
* Participants with high-risk for breast cancer who have received chemopreventive drugs in the past
* Participants with multicentric breast cancer, unless all tumors are HER2+
* Participants with bilateral breast cancer
* Participants who have undergone an excisional biopsy of primary tumor and/or axillary lymph nodes
* Axillary lymph node dissection (ALND) prior to initiation of neoadjuvant therapy
* Sentinel lymph node biopsy (SLNB) prior to neoadjuvant therapy

Exclusion Criterion for Treatment with Adjuvant Trastuzumab Emtansine (Arm E):

* Current Grade ≥3 peripheral neuropathy (according to the NCI CTCAE v5.0)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2025-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (45):
- Argentina (2):
  - Centro de Investigaciones Médicas y Desarrollo LC S.R.L, Buenos Aires, Ciudad Autónoma de BuenosAires
  - Centro Oncologico Korben, Ciudad Autonoma Buenos Aires
- Bosnia and Herzegovina (2):
  - University Clinical Center of the Republic of Srpska, Banja Luka
  - Cantonal Hospital Zenica, Zenica
- Brazil (4):
  - Crio - Centro Regional Integrado de Oncologia, Fortaleza, Ceará
  - Hospital Araujo Jorge, Goiânia, Goiás
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Clinica de Pesquisa e Centro de Estudos em Oncologia Ginecologica e Mamaria Ltda, São Paulo, São Paulo
- Bulgaria (3):
  - Multiprofile Hospital for Active Treatment Uni Hospital, Panagyurishte
  - Complex Oncology Center - Plovdiv First Internal Chemotherapy Department, Plovdiv
  - MHAT Nadezhda, Sofia
- Canada (5):
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - North York General Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - Hopital du Saint Sacrement, Québec, Quebec
- Chile (2):
  - Clinica Vespucio, Santiago
  - Centro de Estudios Clínicos SAGA, Santiago
- Costa Rica (3):
  - Clinica CIMCA, San José
  - ICIMED Instituto de Investigación en Ciencias Médicas, San José
  - Hospital Metropolitano (Sede Lindora-Santa Ana), San José
- Clinical Hospital Centre Zagreb, Zagreb, Croatia
- India (2):
  - Saifee Hospital, Mumbai, Maharashtra
  - TATA Medical Centre, Kolkata, West Bengal
- Kenya (2):
  - International Cancer Institute (ICI), Eldoret
  - The Aga Khan University-Kenya., Nairobi
- Mexico (3):
  - Iem-Fucam, D.F., Mexico City
  - Health Pharma Professional Research, Mexico City, Mexico City
  - Oncologico Potosino, San Luis Potosí City, San Luis Potosí
- Peru (2):
  - Instituto Regional de Enfermedades Neoplásicas del Sur, Arequipa
  - Oncocenter Peru S.A.C., Lima
- Singapore (2):
  - National Cancer Centre, Singapore
  - Tan Tock Seng Hospital, Singapore
- South Africa (2):
  - Medical Oncology Centre of Rosebank, Johannesburg
  - Wilgers Oncology Centre, Pretoria
- South Korea (2):
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (3):
  - Complejo Hospitalario de Jaen-Hospital Universitario Medico Quirurgico, Jaén
  - Hospital Universitario Virgen de Arrixaca, Murcia
  - Hospital Clinico Universitario de Salamanca, Salamanca
- Turkey (Türkiye) (5):
  - Gulhane Training and Research Hospital, Ankara
  - Ankara City Hospital, Ankara
  - Trakya University Medical Faculty Research And Practice Hospital Medical Oncology Department, Edirne
  - Ba?c?lar Medipol Mega Üniversite Hastanesi, Istanbul
  - Hacettepe Uni Medical Faculty Hospital, Sihhiye/Ankara

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 347 participants (1 participant was re-randomized to the same PH FDC SC arm) with early or locally advanced or inflammatory human epidermal growth factor receptor 2-positive (HER2+) breast cancer took part in the study at 45 investigative sites across 17 countries. The study is still ongoing. The health care professionals (HCPs) treating the participants were not enrolled in the study. The HCPs only completed the HCP questionnaire (HCPQ).
Pre-assignment Details: Participants in Neoadjuvant Phase (NP) received either pertuzumab & trastuzumab intravenously (P+H IV) or as a fixed-dose combination, subcutaneously (PH FDC SC), along with chemotherapy. Participants who completed NP, underwent surgical resection & achieved pCR entered Adjuvant Phase to receive PH FDC SC in a run-in period, followed by a cross-over period & then a continuation period at home/hospital. Participants who had residual disease after surgery received trastuzumab emtansine IV.
Groups:
- Arm A, Neoadjuvant Phase: P+H IV: Participants received a loading dose of pertuzumab, 840 milligrams (mg), and trastuzumab, 8 milligrams per kilogram (mg/kg), as an IV infusion on Day 1 of Cycle 1 (Cycle length = 21 days), followed by maintenance doses of pertuzumab, 420 mg and trastuzumab, 6 mg/kg, as an IV infusion, every 3 weeks (Q3W) along with neoadjuvant chemotherapy based on investigator's choice, for 6-8 cycles (depending on the chosen neoadjuvant scheme).
- Arm B, Neoadjuvant Phase: PH FDC SC: Participants received a loading dose of pertuzumab, 1200 mg, trastuzumab, 600 mg, and recombinant human PH20 hyaluronidase (rHuPH20), 30,000 units (U), as a SC injection on Day 1 of Cycle 1 (Cycle length = 21 days) followed by maintenance doses of pertuzumab, 600 mg, trastuzumab, 600 mg and rHuPH20, 20,000 U, as a SC injection, Q3W along with neoadjuvant chemotherapy based on investigator's choice, for 6-8 cycles (depending on the chosen neoadjuvant scheme).
- Adjuvant Run-in Phase: PH FDC SC in Hospital: Participants who achieved pathologic complete response (pCR) after surgery received a loading dose of pertuzumab, 1200 mg, trastuzumab, 600 mg, and rHuPH20, 30,000 U, as a SC injection on Day 1 of Cycle 1 followed by maintenance dose of pertuzumab, 600 mg, trastuzumab, 600 mg and rHuPH20, 20,000 U, as a SC injection, on Day 1 of Cycle 2 (Cycle length = 21 days).
- Arm C, Adjuvant Cross-over Phase: PH FDC SC in Hospital, Then at Home: Participants who completed the run-in period and were randomized to Arm C received maintenance doses of pertuzumab, 600 mg, trastuzumab, 600 mg, and rHuPH20, 20,000 U, as a SC injection for the first 3 cycles in the hospital setting, followed by 3 cycles in the home setting (Cycle length = 21 days).
- Arm D, Adjuvant Cross-Over Phase: PH FDC SC at Home, Then in Hospital: Participants who completed the run-in period and were randomized to Arm D received maintenance doses of pertuzumab, 600 mg, trastuzumab, 600 mg, and rHuPH20, 20,000 U, as a SC injection for the first 3 cycles in the home setting, followed by 3 cycles in the hospital setting (Cycle length = 21 days).
- Arm C, Adjuvant Continuation Phase: PH FDC SC: Participants randomized to Arm C and who completed the cross-over period had an option to receive further treatment in either the home or hospital setting with maintenance doses of pertuzumab, 600 mg, trastuzumab, 600 mg, and rHuPH20, 20,000 U, as a SC injection up to a maximum of 18 cycles (Cycle length = 21 days).
- Arm D, Adjuvant Continuation Phase: PH FDC SC: Participants randomized to Arm D and who completed the cross-over period had an option to receive further treatment in either the home or hospital setting received maintenance doses of pertuzumab, 600 mg, trastuzumab, 600 mg, and rHuPH20, 20,000 U, as a SC injection up to a maximum of 18 cycles (Cycle length = 21 days).
- Arm E, Adjuvant Phase: Trastuzumab Emtansine IV: Participants who did not achieve pCR after surgery received trastuzumab emtansine, 3.6 mg/kg, as an IV infusion for 90 minutes as an initial dose. Thereafter, participants received trastuzumab emtansine, 3.6 mg/kg, as an IV infusion for 30 minutes, Q3W for 14 cycles (Cycle length = 21 days).
Period: Neoadjuvant Phase
Arm/Group | Arm A, Neoadjuvant Phase: P+H IV | Arm B, Neoadjuvant Phase: PH FDC SC | Adjuvant Run-in Phase: PH FDC SC in Hospital | Arm C, Adjuvant Cross-over Phase: PH FDC SC in Hospital, Then at Home | Arm D, Adjuvant Cross-Over Phase: PH FDC SC at Home, Then in Hospital | Arm C, Adjuvant Continuation Phase: PH FDC SC | Arm D, Adjuvant Continuation Phase: PH FDC SC | Arm E, Adjuvant Phase: Trastuzumab Emtansine IV
Started | 116 | 231 | 0 | 0 | 0 | 0 | 0 | 0
Neoadjuvant Safety Analysis Set (SASab) (SASab included all randomized participants who received at least one study treatment during the neoadjuvant phase.) | 115 | 228 | 0 | 0 | 0 | 0 | 0 | 0
Completed Neoadjuvant Treatment | 114 | 210 | 0 | 0 | 0 | 0 | 0 | 0
Completed Surgery | 113 | 207 | 0 | 0 | 0 | 0 | 0 | 0
Continued Into the Run-in Period | 68 | 126 | 0 | 0 | 0 | 0 | 0 | 0
Continued Into Trastuzumab Emtansine IV Arm | 43 | 74 | 0 | 0 | 0 | 0 | 0 | 0
Switched From IV to SC Treatment | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed (Completed Neoadjuvant Treatment and Surgery and Continued to Adjuvant Phase) | 111 | 200 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 5 | 31 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 8 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 11 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Reason not Specified | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Treatment Intolerance | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Adjuvant Phase: Run-in Period
Arm/Group | Arm A, Neoadjuvant Phase: P+H IV | Arm B, Neoadjuvant Phase: PH FDC SC | Adjuvant Run-in Phase: PH FDC SC in Hospital | Arm C, Adjuvant Cross-over Phase: PH FDC SC in Hospital, Then at Home | Arm D, Adjuvant Cross-Over Phase: PH FDC SC at Home, Then in Hospital | Arm C, Adjuvant Continuation Phase: PH FDC SC | Arm D, Adjuvant Continuation Phase: PH FDC SC | Arm E, Adjuvant Phase: Trastuzumab Emtansine IV
Started (Received ≥1 Dose of Adjuvant Run-in Treatment) | 0 | 0 | 194 (All participants that achieved pCR without discontinuing after surgery.) | 0 | 0 | 0 | 0 | 0
Completed (Completed Adjuvant Run-in Treatment) | 0 | 0 | 194 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Adjuvant Phase: Cross-over Period
Arm/Group | Arm A, Neoadjuvant Phase: P+H IV | Arm B, Neoadjuvant Phase: PH FDC SC | Adjuvant Run-in Phase: PH FDC SC in Hospital | Arm C, Adjuvant Cross-over Phase: PH FDC SC in Hospital, Then at Home | Arm D, Adjuvant Cross-Over Phase: PH FDC SC at Home, Then in Hospital | Arm C, Adjuvant Continuation Phase: PH FDC SC | Arm D, Adjuvant Continuation Phase: PH FDC SC | Arm E, Adjuvant Phase: Trastuzumab Emtansine IV
Started (Randomized to Adjuvant Cross-Over Treatment Arms) | 0 | 0 | 0 | 98 (1 participant was randomized but didn't receive any treatment.) | 96 | 0 | 0 | 0
Received ≥1 Dose of Adjuvant Cross-Over Treatment | 0 | 0 | 0 | 97 | 96 | 0 | 0 | 0
Completed (Completed Adjuvant Cross-Over Treatment) | 0 | 0 | 0 | 96 | 93 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Treatment Intolerance | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Adjuvant Phase: Continuation Period
Arm/Group | Arm A, Neoadjuvant Phase: P+H IV | Arm B, Neoadjuvant Phase: PH FDC SC | Adjuvant Run-in Phase: PH FDC SC in Hospital | Arm C, Adjuvant Cross-over Phase: PH FDC SC in Hospital, Then at Home | Arm D, Adjuvant Cross-Over Phase: PH FDC SC at Home, Then in Hospital | Arm C, Adjuvant Continuation Phase: PH FDC SC | Arm D, Adjuvant Continuation Phase: PH FDC SC | Arm E, Adjuvant Phase: Trastuzumab Emtansine IV
Started | 0 | 0 | 0 | 0 | 0 | 96 | 93 (1 participant discontinued after having completed cross-over treatment, and proceeded to follow-up and study completion.) | 0
Chose Home Setting for Continuation Treatment | 0 | 0 | 0 | 0 | 0 | 66 | 50 | 0
Chose Hospital Setting for Continuation Treatment | 0 | 0 | 0 | 0 | 0 | 30 | 42 | 0
Received ≥1 Dose of Continuation Treatment | 0 | 0 | 0 | 0 | 0 | 96 | 89 | 0
Completed (Completed Adjuvant Continuation Treatment) | 0 | 0 | 0 | 0 | 0 | 82 | 81 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 14 | 12 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Non-compliance With Study Drug | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Reason not Specified | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Ongoing in Treatment | 0 | 0 | 0 | 0 | 0 | 11 | 9 | 0
Period: Adjuvant Phase: Trastuzumab Emtansine IV
Arm/Group | Arm A, Neoadjuvant Phase: P+H IV | Arm B, Neoadjuvant Phase: PH FDC SC | Adjuvant Run-in Phase: PH FDC SC in Hospital | Arm C, Adjuvant Cross-over Phase: PH FDC SC in Hospital, Then at Home | Arm D, Adjuvant Cross-Over Phase: PH FDC SC at Home, Then in Hospital | Arm C, Adjuvant Continuation Phase: PH FDC SC | Arm D, Adjuvant Continuation Phase: PH FDC SC | Arm E, Adjuvant Phase: Trastuzumab Emtansine IV
Started (Received ≥1 Dose of Trastuzumab Emtansine) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 117 (All participants that exhibited residual disease after surgery.)
Completed (Completed Trastuzumab Emtansine Treatment) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 77
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 40
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Reason not Specified | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Treatment intolerance | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Not completed — Ongoing in Treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 25
Period: Follow-up Period
Arm/Group | Arm A, Neoadjuvant Phase: P+H IV | Arm B, Neoadjuvant Phase: PH FDC SC | Adjuvant Run-in Phase: PH FDC SC in Hospital | Arm C, Adjuvant Cross-over Phase: PH FDC SC in Hospital, Then at Home | Arm D, Adjuvant Cross-Over Phase: PH FDC SC at Home, Then in Hospital | Arm C, Adjuvant Continuation Phase: PH FDC SC | Arm D, Adjuvant Continuation Phase: PH FDC SC | Arm E, Adjuvant Phase: Trastuzumab Emtansine IV
Started | 0 | 0 | 0 | 0 | 0 | 85 | 87 | 87
Completed | 0 | 0 | 0 | 0 | 0 | 40 | 40 | 34
Not Completed | 0 | 0 | 0 | 0 | 0 | 45 | 47 | 53
Not completed — Ongoing in Follow-up | 0 | 0 | 0 | 0 | 0 | 44 | 45 | 51
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Neoadjuvant full analysis set (FASab) included all randomized participants, regardless of whether they received treatment. The HCPs were not enrolled in this study. Hence, no baseline data were planned to be collected for the HCPs responding to HCPQs.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A, Neoadjuvant Phase: P+H IV | Arm B, Neoadjuvant Phase: PH FDC SC | Total
Number analyzed (Participants) | 116 | 231 | 347
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (11.0) | 52.9 (11.7) | 52.2 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 230 | 346
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 52 | 93 | 145
  Not Hispanic or Latino | 54 | 118 | 172
  Unknown or Not Reported | 10 | 20 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 15 | 35 | 50
  Asian | 12 | 32 | 44
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 10 | 23 | 33
  White | 66 | 123 | 189
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 10 | 13 | 23

OUTCOME MEASURES:

1. Primary Outcome: Cross-over Period: Percentage of Participants Who Preferred the Administration of PH FDC SC in the Home Setting Compared With the Hospital Setting in Question 1 of the Patient Preference Questionnaire (PPQ)
Description: The PPQ was used to evaluate the participant preference for PH FDC SC compared to P+H IV. Participants completed the PPQ, where Question (Q) 1 was: "All things considered, which setting for your treatment did you prefer?" Participants were required to select one of the following options: home, hospital or no preference. The reported results show the percentage of participants who preferred receiving PH FDC SC at home setting over the hospital setting. Percentages were rounded off.
Time Frame: Upon completion of adjuvant cross-over period (Day 1 of Cycle 8 or 9; Cycle length = 21 days)
Population: Adjuvant cross-over modified intent-to-treat (mITTcross) population included all randomized participants assigned into the cross-over period who received at least one dose of PH FDC SC, completed Question 1 of the PPQ, and completed radiotherapy before entering the cross-over period.
Measure: Number; unit: percentage of participants
Arm/Group | Arm C, Adjuvant Cross-over Phase: PH FDC SC in Hospital, Then at Home | Arm D, Adjuvant Cross-Over Phase: PH FDC SC at Home, Then in Hospital
Number analyzed (Participants) | 87 | 83
percentage of participants
  Home | 69.0 | 59.0
  Hospital | 23.0 | 39.8
  No Preference | 8.0 | 1.2

2. Secondary Outcome: Neoadjuvant Phase: Percentage of HCPs by Their Responses to Question 1a of HCPQ - Drug Preparation Area
Description: HCP was defined as any personnel involved in the drug preparation and/or drug administration processes. HCPs who have had experience with preparation of P+H IV and/or administration of PH FDC SC completed the following question of the HCPQ: Q1a: "Please indicate which treatment preparation the estimates relate to". HCPs were required to select one of the following options: PH FDC SC or P+H IV. The response to Q1a was used to further assess Q1b: How long did it take to prepare the treatment for use? Percentages were rounded off.
Time Frame: Day 1 of Cycles 1-8 (Cycle length = 21 days)
Population: Participants could have changed from P+H IV treatment to PH FDC SC treatment, in exceptional circumstances and at the investigator discretion. Overall number analyzed is the number of HCPs who answered Q1a of the HCPQ. Number analyzed is the number of HCPs who answered Q1a of the HCPQ at the specified time point.
Measure: Number; unit: percentage of HCPs
Arm/Group | Arm A, Neoadjuvant Phase: P+H IV | Arm B, Neoadjuvant Phase: PH FDC SC
Number analyzed (Participants) | 113 | 211
percentage of HCPs
  Cycle 1 Day 1: PH FDC SC: number analyzed (Participants) | 62 | 121
  Cycle 1 Day 1: PH FDC SC | 0 | 100
  Cycle 1 Day 1: P+H IV: number analyzed (Participants) | 62 | 121
  Cycle 1 Day 1: P+H IV | 100 | 0
  Cycle 2 Day 1: PH FDC SC: number analyzed (Participants) | 62 | 116
  Cycle 2 Day 1: PH FDC SC | 0 | 100
  Cycle 2 Day 1: P+H IV: number analyzed (Participants) | 62 | 116
  Cycle 2 Day 1: P+H IV | 100 | 0
  Cycle 3 Day 1: PH FDC SC: number analyzed (Participants) | 62 | 114
  Cycle 3 Day 1: PH FDC SC | 0 | 100
  Cycle 3 Day 1: P+H IV: number analyzed (Participants) | 62 | 114
  Cycle 3 Day 1: P+H IV | 100 | 0
  Cycle 4 Day 1: PH FDC SC: number analyzed (Participants) | 62 | 114
  Cycle 4 Day 1: PH FDC SC | 1.6 | 100
  Cycle 4 Day 1: P+H IV: number analyzed (Participants) | 62 | 114
  Cycle 4 Day 1: P+H IV | 98.4 | 0
  Cycle 5 Day 1: PH FDC SC | 0.9 | 100
  Cycle 5 Day 1: P+H IV | 99.1 | 0
  Cycle 6 Day 1: PH FDC SC: number analyzed (Participants) | 112 | 207
  Cycle 6 Day 1: PH FDC SC | 0.9 | 100
  Cycle 6 Day 1: P+H IV: number analyzed (Participants) | 112 | 207
  Cycle 6 Day 1: P+H IV | 99.1 | 0
  Cycle 7 Day 1: PH FDC SC: number analyzed (Participants) | 58 | 111
  Cycle 7 Day 1: PH FDC SC | 0 | 100
  Cycle 7 Day 1: P+H IV: number analyzed (Participants) | 58 | 111
  Cycle 7 Day 1: P+H IV | 100 | 0
  Cycle 8 Day 1: PH FDC SC: number analyzed (Participants) | 56 | 107
  Cycle 8 Day 1: PH FDC SC | 0 | 100
  Cycle 8 Day 1: P+H IV: number analyzed (Participants) | 56 | 107
  Cycle 8 Day 1: P+H IV | 100 | 0

3. Secondary Outcome: Neoadjuvant Phase: Duration of Treatment Preparation, According to Healthcare Professionals' Responses to Question 1b of HCPQ - Drug Preparation Area
Description: HCP was defined as any personnel involved in the drug preparation and/or drug administration processes. HCPs who have had experience with preparation of P+H IV and/or administration of PH FDC SC completed the following question of the HCPQ: Q1b: "How long did it take to prepare the treatment for use?" This was a follow up question to Q1a: "Please indicate which treatment preparation the estimates relate to" for which HCPs were required to select one of the following options: PH FDC SC or P+H IV.
Time Frame: Day 1 of Cycles 1-8 (Cycle length = 21 days)
Population: Overall number analyzed is the number of HCPs who answered Q1b of the HCPQ. Number analyzed is the number of HCPs who answered Q1b of the HCPQ at the specified time point.
Measure: Median (Full Range); unit: minutes
Arm/Group | Arm A, Neoadjuvant Phase: P+H IV | Arm B, Neoadjuvant Phase: PH FDC SC
Number analyzed (Participants) | 113 | 211
minutes
  Cycle 1 Day 1: number analyzed (Participants) | 62 | 120
  Cycle 1 Day 1 | 20.0 [1 to 120] | 5.0 [0 to 30]
  Cycle 2 Day 1: number analyzed (Participants) | 62 | 115
  Cycle 2 Day 1 | 20.5 [1 to 50] | 5.0 [0 to 40]
  Cycle 3 Day 1: number analyzed (Participants) | 62 | 113
  Cycle 3 Day 1 | 20.0 [1 to 50] | 5.0 [1 to 35]
  Cycle 4 Day 1: number analyzed (Participants) | 62 | 113
  Cycle 4 Day 1 | 20.0 [1 to 50] | 5.0 [1 to 30]
  Cycle 5 Day 1 | 20.0 [1 to 110] | 5.0 [1 to 52]
  Cycle 6 Day 1: number analyzed (Participants) | 112 | 207
  Cycle 6 Day 1 | 20.0 [1 to 410] | 5.0 [1 to 131]
  Cycle 7 Day 1: number analyzed (Participants) | 58 | 111
  Cycle 7 Day 1 | 13.5 [4 to 90] | 4.0 [1 to 45]
  Cycle 8 Day 1: number analyzed (Participants) | 56 | 106
  Cycle 8 Day 1 | 15.0 [4 to 90] | 5.0 [1 to 45]

4. Secondary Outcome: Neoadjuvant Phase: Percentage of HCPs by Their Response to Question 2 of the HCPQ - Drug Preparation Area
Description: HCP=any personnel involved in the drug preparation and/or drug administration processes. HCPs who have had experience with preparation of P+H IV and/or administration of PH FDC SC completed the following question 2 of the HCPQs: In your opinion, if all P+H IV infusions were switched to PH FDC SC injections, please indicate how strongly you agree/disagree with each of the following statements. 2a: Staff will have increased availability for other tasks in the pharmacy. 2b: Administrative procedures related to PH FDC SC require less time. 2c: Using PH FDC SC provides more flexibility for pharmacy staff in managing their workload. 2d: As PH FDC SC is fixed-dose, potential dosing errors are avoided. 2e: As PH FDC SC is fixed-dose, there is less drug wastage. 2f: Less storage space for PH FDC SC-related supplies is required in the pharmacy, as there is no need for reconstitution. 2g: Number of preparation steps & staff time commitment are reduced. Percentages were rounded off.
Time Frame: Up to Day 1 of Cycle 8 (Cycle length = 21 days)
Population: Overall number analyzed is the number of HCPs who answered Q2 of the HCPQ. Number analyzed is the number of HCPs who responded to each sub-question of Q2 (Q2a-Q2g) of the HCPQ.
Measure: Number; unit: percentage of HCPs
Arm/Group | Arm A, Neoadjuvant Phase: P+H IV | Arm B, Neoadjuvant Phase: PH FDC SC
Number analyzed (Participants) | 89 | 165
percentage of HCPs
  Q2a: Strongly Disagree: number analyzed (Participants) | 89 | 164
  Q2a: Strongly Disagree | 1.1 | 2.4
  Q2a: Disagree: number analyzed (Participants) | 89 | 164
  Q2a: Disagree | 3.4 | 2.4
  Q2a: Neutral: number analyzed (Participants) | 89 | 164
  Q2a: Neutral | 13.5 | 11.0
  Q2a: Agree: number analyzed (Participants) | 89 | 164
  Q2a: Agree | 25.8 | 38.4
  Q2a: Strongly Agree: number analyzed (Participants) | 89 | 164
  Q2a: Strongly Agree | 52.8 | 39.6
  Q2a: Not Applicable: number analyzed (Participants) | 89 | 164
  Q2a: Not Applicable | 3.4 | 6.1
  Q2b: Strongly Disagree: number analyzed (Participants) | 89 | 164
  Q2b: Strongly Disagree | 4.5 | 2.4
  Q2b: Disagree: number analyzed (Participants) | 89 | 164
  Q2b: Disagree | 12.4 | 15.2
  Q2b: Neutral: number analyzed (Participants) | 89 | 164
  Q2b: Neutral | 13.5 | 14.6
  Q2b: Agree: number analyzed (Participants) | 89 | 164
  Q2b: Agree | 18.0 | 25.6
  Q2b: Strongly Agree: number analyzed (Participants) | 89 | 164
  Q2b: Strongly Agree | 47.2 | 35.4
  Q2b: Not Applicable: number analyzed (Participants) | 89 | 164
  Q2b: Not Applicable | 4.5 | 6.7
  Q2c: Strongly Disagree: number analyzed (Participants) | 89 | 164
  Q2c: Strongly Disagree | 1.1 | 1.2
  Q2c: Disagree: number analyzed (Participants) | 89 | 164
  Q2c: Disagree | 4.5 | 2.4
  Q2c: Neutral: number analyzed (Participants) | 89 | 164
  Q2c: Neutral | 11.2 | 14.0
  Q2c: Agree: number analyzed (Participants) | 89 | 164
  Q2c: Agree | 28.1 | 41.5
  Q2c: Strongly Agree: number analyzed (Participants) | 89 | 164
  Q2c: Strongly Agree | 50.6 | 34.1
  Q2c: Not Applicable: number analyzed (Participants) | 89 | 164
  Q2c: Not Applicable | 4.5 | 6.7
  Q2d: Strongly Disagree: number analyzed (Participants) | 89 | 164
  Q2d: Strongly Disagree | 1.1 | 1.2
  Q2d: Disagree: number analyzed (Participants) | 89 | 164
  Q2d: Disagree | 2.2 | 2.4
  Q2d: Neutral: number analyzed (Participants) | 89 | 164
  Q2d: Neutral | 2.2 | 7.9
  Q2d: Agree: number analyzed (Participants) | 89 | 164
  Q2d: Agree | 28.1 | 36.0
  Q2d: Strongly Agree: number analyzed (Participants) | 89 | 164
  Q2d: Strongly Agree | 61.8 | 46.3
  Q2d: Not Applicable: number analyzed (Participants) | 89 | 164
  Q2d: Not Applicable | 4.5 | 6.1
  Q2e: Strongly Disagree: number analyzed (Participants) | 89 | 164
  Q2e: Strongly Disagree | 1.1 | 1.2
  Q2e: Disagree: number analyzed (Participants) | 89 | 164
  Q2e: Disagree | 3.4 | 3.7
  Q2e: Neutral: number analyzed (Participants) | 89 | 164
  Q2e: Neutral | 1.1 | 6.1
  Q2e: Strongly Agree: number analyzed (Participants) | 89 | 164
  Q2e: Strongly Agree | 31.5 | 35.4
  Q2e: Agree: number analyzed (Participants) | 89 | 164
  Q2e: Agree | 58.4 | 47.6
  Q2e: Not Available: number analyzed (Participants) | 89 | 164
  Q2e: Not Available | 4.5 | 6.1
  Q2f: Strongly Disagree: number analyzed (Participants) | 89 | 164
  Q2f: Strongly Disagree | 1.1 | 1.2
  Q2f: Disagree: number analyzed (Participants) | 89 | 164
  Q2f: Disagree | 5.6 | 6.1
  Q2f: Neutral: number analyzed (Participants) | 89 | 164
  Q2f: Neutral | 10.1 | 12.2
  Q2f: Strongly Agree: number analyzed (Participants) | 89 | 164
  Q2f: Strongly Agree | 24.7 | 33.5
  Q2f: Agree: number analyzed (Participants) | 89 | 164
  Q2f: Agree | 53.9 | 40.9
  Q2f: Not available: number analyzed (Participants) | 89 | 164
  Q2f: Not available | 4.5 | 6.1
  Q2g: Strongly Disagree | 1.1 | 1.8
  Q2g: Disagree | 7.9 | 4.2
  Q2g: Neutral | 7.9 | 6.1
  Q2g: Strongly Agree | 23.6 | 36.4
  Q2g: Agree | 56.2 | 44.8
  Q2g: Not available | 3.4 | 6.7

5. Secondary Outcome: Neoadjuvant Phase: Percentage of HCPs by Their Responses to Questions 1a-1e of the HCPQ - Administering Treatment
Description: HCP was defined as any personnel involved in the drug preparation and/or drug administration processes. HCPs who have had experience with administration of P+H IV and/or PH FDC SC completed the following Questions of the HCPQ: Q1a: Please indicate which treatment preparation the estimates relate to. Q1b: Did the participant have existing IV access? Q1c: If new IV access was needed for this cycle of treatment, please indicate what type of IV access was provided. Q1d: What type of existing IV access did the participant have? Q1e: When did the existing IV access place? Percentages were rounded off.
  PICC = peripherally inserted central catheter.
Time Frame: Day 1 of Cycles 1-8 (Cycle length = 21 days)
Population: Participants could have changed from P+H IV treatment to PH FDC SC treatment, in exceptional circumstances and at the investigator discretion. Overall number analyzed is the number of HCPs who answered Q1a to Q1e of the HCPQ. Number analyzed is the number of HCPs who answered Q1a to Q1e of the HCPQ at the specified time point.
Measure: Number; unit: percentage of HCPs
Arm/Group | Arm A, Neoadjuvant Phase: P+H IV | Arm B, Neoadjuvant Phase: PH FDC SC
Number analyzed (Participants) | 112 | 213
percentage of HCPs
  Cycle 1 Day 1: Q1a: PH FDC SC: number analyzed (Participants) | 63 | 122
  Cycle 1 Day 1: Q1a: PH FDC SC | 0 | 100
  Cycle 1 Day 1: Q1a: P+H IV: number analyzed (Participants) | 63 | 122
  Cycle 1 Day 1: Q1a: P+H IV | 100 | 0
  Cycle 1 Day 1: Q1b: Yes: number analyzed (Participants) | 62 | 1
  Cycle 1 Day 1: Q1b: Yes | 24.2 | 0
  Cycle 1 Day 1: Q1b: No: number analyzed (Participants) | 62 | 1
  Cycle 1 Day 1: Q1b: No | 75.8 | 100
  Cycle 1 Day 1: Q1c: Peripheral Vein Cannulation: number analyzed (Participants) | 43 | 7
  Cycle 1 Day 1: Q1c: Peripheral Vein Cannulation | 90.7 | 100
  Cycle 1 Day 1: Q1c: PICC: number analyzed (Participants) | 43 | 7
  Cycle 1 Day 1: Q1c: PICC | 0 | 0
  Cycle 1 Day 1: Q1c: Central Venous Catheter: number analyzed (Participants) | 43 | 7
  Cycle 1 Day 1: Q1c: Central Venous Catheter | 9.3 | 0
  Cycle 1 Day 1: Q1d: Central Venous Catheter: number analyzed (Participants) | 15 | 2
  Cycle 1 Day 1: Q1d: Central Venous Catheter | 40.0 | 0
  Cycle 1 Day 1: Q1d: PICC: number analyzed (Participants) | 15 | 2
  Cycle 1 Day 1: Q1d: PICC | 33.3 | 50.0
  Cycle 1 Day 1: Q1d: Port-a-Cath: number analyzed (Participants) | 15 | 2
  Cycle 1 Day 1: Q1d: Port-a-Cath | 26.7 | 50.0
  Cycle 1 Day 1: Q1d: Tunneled Central Venous Catheter: number analyzed (Participants) | 15 | 2
  Cycle 1 Day 1: Q1d: Tunneled Central Venous Catheter | 0 | 0
  Cycle 1 Day 1: Q1e: Within 7 Days Prior Today: number analyzed (Participants) | 6 | 6
  Cycle 1 Day 1: Q1e: Within 7 Days Prior Today | 50.0 | 16.7
  Cycle 1 Day 1: Q1e: > 7 < 14 Days Prior Today: number analyzed (Participants) | 6 | 6
  Cycle 1 Day 1: Q1e: > 7 < 14 Days Prior Today | 0 | 33.3
  Cycle 1 Day 1: Q1e: > 14 < 30 Days Prior Today: number analyzed (Participants) | 6 | 6
  Cycle 1 Day 1: Q1e: > 14 < 30 Days Prior Today | 0 | 0
  Cycle 1 Day 1: Q1e: Other: number analyzed (Participants) | 6 | 6
  Cycle 1 Day 1: Q1e: Other | 50.0 | 50.0
  Cycle 2 Day 1: Q1a: PH FDC SC: number analyzed (Participants) | 62 | 118
  Cycle 2 Day 1: Q1a: PH FDC SC | 0 | 100
  Cycle 2 Day 1: Q1a: P+H IV: number analyzed (Participants) | 62 | 118
  Cycle 2 Day 1: Q1a: P+H IV | 100 | 0
  Cycle 2 Day 1: Q1b: Yes: number analyzed (Participants) | 61 | 5
  Cycle 2 Day 1: Q1b: Yes | 23.0 | 60.0
  Cycle 2 Day 1: Q1b: No: number analyzed (Participants) | 61 | 5
  Cycle 2 Day 1: Q1b: No | 77.0 | 40.0
  Cycle 2 Day 1: Q1c: Peripheral Vein Cannulation: number analyzed (Participants) | 44 | 3
  Cycle 2 Day 1: Q1c: Peripheral Vein Cannulation | 88.6 | 66.7
  Cycle 2 Day 1: Q1c: PICC: number analyzed (Participants) | 44 | 3
  Cycle 2 Day 1: Q1c: PICC | 0 | 0
  Cycle 2 Day 1: Q1c: Central Venous Catheter: number analyzed (Participants) | 44 | 3
  Cycle 2 Day 1: Q1c: Central Venous Catheter | 11.4 | 33.3
  Cycle 2 Day 1: Q1d: Central Venous Catheter: number analyzed (Participants) | 14 | 5
  Cycle 2 Day 1: Q1d: Central Venous Catheter | 35.7 | 40.0
  Cycle 2 Day 1: Q1d: PICC: number analyzed (Participants) | 14 | 5
  Cycle 2 Day 1: Q1d: PICC | 28.6 | 20.0
  Cycle 2 Day 1: Q1d: Port-a-Cath: number analyzed (Participants) | 14 | 5
  Cycle 2 Day 1: Q1d: Port-a-Cath | 35.7 | 40.0
  Cycle 2 Day 1: Q1d: Tunneled Central Venous Catheter: number analyzed (Participants) | 14 | 5
  Cycle 2 Day 1: Q1d: Tunneled Central Venous Catheter | 0 | 0
  Cycle 2 Day 1: Q1e: Within 7 Days Prior Today: number analyzed (Participants) | 6 | 8
  Cycle 2 Day 1: Q1e: Within 7 Days Prior Today | 0 | 0
  Cycle 2 Day 1: Q1e: > 7 < 14 Days Prior Today: number analyzed (Participants) | 6 | 8
  Cycle 2 Day 1: Q1e: > 7 < 14 Days Prior Today | 0 | 0
  Cycle 2 Day 1: Q1e: > 14 < 30 Days Prior Today: number analyzed (Participants) | 6 | 8
  Cycle 2 Day 1: Q1e: > 14 < 30 Days Prior Today | 16.7 | 62.5
  Cycle 2 Day 1: Q1e: Other: number analyzed (Participants) | 6 | 8
  Cycle 2 Day 1: Q1e: Other | 83.3 | 37.5
  Cycle 3 Day 1: Q1a: PH FDC SC: number analyzed (Participants) | 61 | 113
  Cycle 3 Day 1: Q1a: PH FDC SC | 0 | 100
  Cycle 3 Day 1: Q1a: P+H IV: number analyzed (Participants) | 61 | 113
  Cycle 3 Day 1: Q1a: P+H IV | 100 | 0
  Cycle 3 Day 1: Q1b: Yes: number analyzed (Participants) | 61 | 3
  Cycle 3 Day 1: Q1b: Yes | 26.2 | 100
  Cycle 3 Day 1: Q1b: No: number analyzed (Participants) | 61 | 3
  Cycle 3 Day 1: Q1b: No | 73.8 | 0
  Cycle 3 Day 1: Q1c: Peripheral Vein Cannulation: number analyzed (Participants) | 42 | 4
  Cycle 3 Day 1: Q1c: Peripheral Vein Cannulation | 88.1 | 100
  Cycle 3 Day 1: Q1c: PICC: number analyzed (Participants) | 42 | 4
  Cycle 3 Day 1: Q1c: PICC | 2.4 | 0
  Cycle 3 Day 1: Q1c: Central Venous Catheter: number analyzed (Participants) | 42 | 4
  Cycle 3 Day 1: Q1c: Central Venous Catheter | 9.5 | 0
  Cycle 3 Day 1: Q1d: Central Venous Catheter: number analyzed (Participants) | 15 | 7
  Cycle 3 Day 1: Q1d: Central Venous Catheter | 33.3 | 57.1
  Cycle 3 Day 1: Q1d: PICC: number analyzed (Participants) | 15 | 7
  Cycle 3 Day 1: Q1d: PICC | 33.3 | 28.6
  Cycle 3 Day 1: Q1d: Port-a-Cath: number analyzed (Participants) | 15 | 7
  Cycle 3 Day 1: Q1d: Port-a-Cath | 33.3 | 14.3
  Cycle 3 Day 1: Q1d: Tunneled Central Venous Catheter: number analyzed (Participants) | 15 | 7
  Cycle 3 Day 1: Q1d: Tunneled Central Venous Catheter | 0 | 0
  Cycle 3 Day 1: Q1e: Within 7 Days Prior Today: number analyzed (Participants) | 6 | 12
  Cycle 3 Day 1: Q1e: Within 7 Days Prior Today | 16.7 | 16.7
  Cycle 3 Day 1: Q1e: > 7 < 14 Days Prior Today: number analyzed (Participants) | 6 | 12
  Cycle 3 Day 1: Q1e: > 7 < 14 Days Prior Today | 0 | 8.3
  Cycle 3 Day 1: Q1e: > 14 < 30 Days Prior Today: number analyzed (Participants) | 6 | 12
  Cycle 3 Day 1: Q1e: > 14 < 30 Days Prior Today | 0 | 25.0
  Cycle 3 Day 1: Q1e: Other: number analyzed (Participants) | 6 | 12
  Cycle 3 Day 1: Q1e: Other | 83.3 | 50.0
  Cycle 4 Day 1: Q1a: PH FDC SC: number analyzed (Participants) | 62 | 113
  Cycle 4 Day 1: Q1a: PH FDC SC | 1.6 | 100
  Cycle 4 Day 1: Q1a: P+H IV: number analyzed (Participants) | 62 | 113
  Cycle 4 Day 1: Q1a: P+H IV | 98.4 | 0
  Cycle 4 Day 1: Q1b: Yes: number analyzed (Participants) | 59 | 2
  Cycle 4 Day 1: Q1b: Yes | 32.2 | 50.0
  Cycle 4 Day 1: Q1b: No: number analyzed (Participants) | 59 | 2
  Cycle 4 Day 1: Q1b: No | 67.8 | 50.0
  Cycle 4 Day 1: Q1c: Peripheral Vein Cannulation: number analyzed (Participants) | 39 | 2
  Cycle 4 Day 1: Q1c: Peripheral Vein Cannulation | 89.7 | 50.0
  Cycle 4 Day 1: Q1c: PICC: number analyzed (Participants) | 39 | 2
  Cycle 4 Day 1: Q1c: PICC | 0 | 0
  Cycle 4 Day 1: Q1c: Central Venous Catheter: number analyzed (Participants) | 39 | 2
  Cycle 4 Day 1: Q1c: Central Venous Catheter | 10.3 | 50.0
  Cycle 4 Day 1: Q1d: Central Venous Catheter: number analyzed (Participants) | 20 | 4
  Cycle 4 Day 1: Q1d: Central Venous Catheter | 30.0 | 50.0
  Cycle 4 Day 1: Q1d: PICC: number analyzed (Participants) | 20 | 4
  Cycle 4 Day 1: Q1d: PICC | 35.0 | 0
  Cycle 4 Day 1: Q1d: Port-a-Cath: number analyzed (Participants) | 20 | 4
  Cycle 4 Day 1: Q1d: Port-a-Cath | 35.0 | 50.0
  Cycle 4 Day 1: Q1d: Tunneled Central Venous Catheter: number analyzed (Participants) | 20 | 4
  Cycle 4 Day 1: Q1d: Tunneled Central Venous Catheter | 0 | 0
  Cycle 4 Day 1: Q1e: Within 7 Days Prior Today: number analyzed (Participants) | 7 | 13
  Cycle 4 Day 1: Q1e: Within 7 Days Prior Today | 0 | 7.7
  Cycle 4 Day 1: Q1e: > 7 < 14 Days Prior Today: number analyzed (Participants) | 7 | 13
  Cycle 4 Day 1: Q1e: > 7 < 14 Days Prior Today | 0 | 0
  Cycle 4 Day 1: Q1e: > 14 < 30 Days Prior Today: number analyzed (Participants) | 7 | 13
  Cycle 4 Day 1: Q1e: > 14 < 30 Days Prior Today | 14.3 | 38.5
  Cycle 4 Day 1: Q1e: Other: number analyzed (Participants) | 7 | 13
  Cycle 4 Day 1: Q1e: Other | 85.7 | 53.8
  Cycle 5 Day 1: Q1a: PH FDC SC | 0.9 | 100
  Cycle 5 Day 1: Q1a: P+H IV | 99.1 | 0
  Cycle 5 Day 1: Q1b: Yes: number analyzed (Participants) | 108 | 4
  Cycle 5 Day 1: Q1b: Yes | 33.3 | 25.0
  Cycle 5 Day 1: Q1b: No: number analyzed (Participants) | 108 | 4
  Cycle 5 Day 1: Q1b: No | 66.7 | 75.0
  Cycle 5 Day 1: Q1c: Port-a-cath: number analyzed (Participants) | 73 | 6
  Cycle 5 Day 1: Q1c: Port-a-cath | 1.4 | 0
  Cycle 5 Day 1: Q1c: Peripheral Vein Cannulation: number analyzed (Participants) | 73 | 6
  Cycle 5 Day 1: Q1c: Peripheral Vein Cannulation | 93.2 | 83.3
  Cycle 5 Day 1: Q1c: PICC: number analyzed (Participants) | 73 | 6
  Cycle 5 Day 1: Q1c: PICC | 0 | 0
  Cycle 5 Day 1: Q1c: Central Venous Catheter: number analyzed (Participants) | 73 | 6
  Cycle 5 Day 1: Q1c: Central Venous Catheter | 5.5 | 16.7
  Cycle 5 Day 1: Q1d: Central Venous Catheter: number analyzed (Participants) | 36 | 6
  Cycle 5 Day 1: Q1d: Central Venous Catheter | 19.4 | 16.7
  Cycle 5 Day 1: Q1d: PICC: number analyzed (Participants) | 36 | 6
  Cycle 5 Day 1: Q1d: PICC | 41.7 | 0
  Cycle 5 Day 1: Q1d: Port-a-Cath: number analyzed (Participants) | 36 | 6
  Cycle 5 Day 1: Q1d: Port-a-Cath | 33.3 | 83.3
  Cycle 5 Day 1: Q1d: Tunneled Central Venous Catheter: number analyzed (Participants) | 36 | 6
  Cycle 5 Day 1: Q1d: Tunneled Central Venous Catheter | 5.6 | 0
  Cycle 5 Day 1: Q1e: Within 7 Days Prior Today: number analyzed (Participants) | 19 | 27
  Cycle 5 Day 1: Q1e: Within 7 Days Prior Today | 21.1 | 7.4
  Cycle 5 Day 1: Q1e: > 7 < 14 Days Prior Today: number analyzed (Participants) | 19 | 27
  Cycle 5 Day 1: Q1e: > 7 < 14 Days Prior Today | 10.5 | 11.1
  Cycle 5 Day 1: Q1e: > 14 < 30 Days Prior Today: number analyzed (Participants) | 19 | 27
  Cycle 5 Day 1: Q1e: > 14 < 30 Days Prior Today | 15.8 | 29.6
  Cycle 5 Day 1: Q1e: Other: number analyzed (Participants) | 19 | 27
  Cycle 5 Day 1: Q1e: Other | 52.6 | 51.9
  Cycle 6 Day 1: Q1a: PH FDC SC: number analyzed (Participants) | 111 | 205
  Cycle 6 Day 1: Q1a: PH FDC SC | 0.9 | 100
  Cycle 6 Day 1: Q1a: P+H IV: number analyzed (Participants) | 111 | 205
  Cycle 6 Day 1: Q1a: P+H IV | 99.1 | 0
  Cycle 6 Day 1: Q1b: Yes: number analyzed (Participants) | 109 | 5
  Cycle 6 Day 1: Q1b: Yes | 34.9 | 40.0
  Cycle 6 Day 1: Q1b: No: number analyzed (Participants) | 109 | 5
  Cycle 6 Day 1: Q1b: No | 65.1 | 60.0
  Cycle 6 Day 1: Q1c: Port-a-cath: number analyzed (Participants) | 72 | 6
  Cycle 6 Day 1: Q1c: Port-a-cath | 2.8 | 0
  Cycle 6 Day 1: Q1c: Peripheral Vein Cannulation: number analyzed (Participants) | 72 | 6
  Cycle 6 Day 1: Q1c: Peripheral Vein Cannulation | 94.4 | 100
  Cycle 6 Day 1: Q1c: PICC: number analyzed (Participants) | 72 | 6
  Cycle 6 Day 1: Q1c: PICC | 0 | 0
  Cycle 6 Day 1: Q1c: Central Venous Catheter: number analyzed (Participants) | 72 | 6
  Cycle 6 Day 1: Q1c: Central Venous Catheter | 2.8 | 0
  Cycle 6 Day 1: Q1d: Central Venous Catheter: number analyzed (Participants) | 37 | 7
  Cycle 6 Day 1: Q1d: Central Venous Catheter | 16.2 | 0
  Cycle 6 Day 1: Q1d: PICC: number analyzed (Participants) | 37 | 7
  Cycle 6 Day 1: Q1d: PICC | 43.2 | 14.3
  Cycle 6 Day 1: Q1d: Port-a-Cath: number analyzed (Participants) | 37 | 7
  Cycle 6 Day 1: Q1d: Port-a-Cath | 32.4 | 85.7
  Cycle 6 Day 1: Q1d: Tunneled Central Venous Catheter: number analyzed (Participants) | 37 | 7
  Cycle 6 Day 1: Q1d: Tunneled Central Venous Catheter | 8.1 | 0
  Cycle 6 Day 1: Q1e: Within 7 Days Prior Today: number analyzed (Participants) | 20 | 31
  Cycle 6 Day 1: Q1e: Within 7 Days Prior Today | 25.0 | 6.5
  Cycle 6 Day 1: Q1e: > 7 < 14 Days Prior Today: number analyzed (Participants) | 20 | 31
  Cycle 6 Day 1: Q1e: > 7 < 14 Days Prior Today | 0 | 9.7
  Cycle 6 Day 1: Q1e: > 14 < 30 Days Prior Today: number analyzed (Participants) | 20 | 31
  Cycle 6 Day 1: Q1e: > 14 < 30 Days Prior Today | 15.0 | 29.0
  Cycle 6 Day 1: Q1e: Other: number analyzed (Participants) | 20 | 31
  Cycle 6 Day 1: Q1e: Other | 60.0 | 54.8
  Cycle 7 Day 1: Q1a: PH FDC SC: number analyzed (Participants) | 57 | 111
  Cycle 7 Day 1: Q1a: PH FDC SC | 0 | 100
  Cycle 7 Day 1: Q1a: P+H IV: number analyzed (Participants) | 57 | 111
  Cycle 7 Day 1: Q1a: P+H IV | 100 | 0
  Cycle 7 Day 1: Q1b: Yes: number analyzed (Participants) | 57 | 3
  Cycle 7 Day 1: Q1b: Yes | 28.1 | 66.7
  Cycle 7 Day 1: Q1b: No: number analyzed (Participants) | 57 | 3
  Cycle 7 Day 1: Q1b: No | 71.9 | 33.3
  Cycle 7 Day 1: Q1c: Peripheral Vein Cannulation: number analyzed (Participants) | 41 | 2
  Cycle 7 Day 1: Q1c: Peripheral Vein Cannulation | 97.6 | 50.0
  Cycle 7 Day 1: Q1c: PICC: number analyzed (Participants) | 41 | 2
  Cycle 7 Day 1: Q1c: PICC | 0 | 0
  Cycle 7 Day 1: Q1c: Central Venous Catheter: number analyzed (Participants) | 41 | 2
  Cycle 7 Day 1: Q1c: Central Venous Catheter | 2.4 | 50.0
  Cycle 7 Day 1: Q1d: Central Venous Catheter: number analyzed (Participants) | 16 | 5
  Cycle 7 Day 1: Q1d: Central Venous Catheter | 6.3 | 0
  Cycle 7 Day 1: Q1d: PICC: number analyzed (Participants) | 16 | 5
  Cycle 7 Day 1: Q1d: PICC | 50.0 | 20.0
  Cycle 7 Day 1: Q1d: Port-a-Cath: number analyzed (Participants) | 16 | 5
  Cycle 7 Day 1: Q1d: Port-a-Cath | 25.0 | 80.0
  Cycle 7 Day 1: Q1d: Tunneled Central Venous Catheter: number analyzed (Participants) | 16 | 5
  Cycle 7 Day 1: Q1d: Tunneled Central Venous Catheter | 18.8 | 0
  Cycle 7 Day 1: Q1e: Within 7 Days Prior Today: number analyzed (Participants) | 13 | 17
  Cycle 7 Day 1: Q1e: Within 7 Days Prior Today | 38.5 | 11.8
  Cycle 7 Day 1: Q1e: > 7 < 14 Days Prior Today: number analyzed (Participants) | 13 | 17
  Cycle 7 Day 1: Q1e: > 7 < 14 Days Prior Today | 0 | 17.6
  Cycle 7 Day 1: Q1e: > 14 < 30 Days Prior Today: number analyzed (Participants) | 13 | 17
  Cycle 7 Day 1: Q1e: > 14 < 30 Days Prior Today | 15.4 | 5.9
  Cycle 7 Day 1: Q1e: Other: number analyzed (Participants) | 13 | 17
  Cycle 7 Day 1: Q1e: Other | 46.2 | 64.7
  Cycle 8 Day 1: Q1a: PH FDC SC: number analyzed (Participants) | 57 | 108
  Cycle 8 Day 1: Q1a: PH FDC SC | 0 | 100
  Cycle 8 Day 1: Q1a: P+H IV: number analyzed (Participants) | 57 | 108
  Cycle 8 Day 1: Q1a: P+H IV | 100 | 0
  Cycle 8 Day 1: Q1b: Yes: number analyzed (Participants) | 57 | 4
  Cycle 8 Day 1: Q1b: Yes | 33.3 | 0
  Cycle 8 Day 1: Q1b: No: number analyzed (Participants) | 57 | 4
  Cycle 8 Day 1: Q1b: No | 66.7 | 100
  Cycle 8 Day 1: Q1c: Peripheral Vein Cannulation: number analyzed (Participants) | 38 | 5
  Cycle 8 Day 1: Q1c: Peripheral Vein Cannulation | 97.4 | 100
  Cycle 8 Day 1: Q1c: PICC: number analyzed (Participants) | 38 | 5
  Cycle 8 Day 1: Q1c: PICC | 0 | 0
  Cycle 8 Day 1: Q1c: Central Venous Catheter: number analyzed (Participants) | 38 | 5
  Cycle 8 Day 1: Q1c: Central Venous Catheter | 2.6 | 0
  Cycle 8 Day 1: Q1d: Central Venous Catheter: number analyzed (Participants) | 19 | 1
  Cycle 8 Day 1: Q1d: Central Venous Catheter | 10.5 | 0
  Cycle 8 Day 1: Q1d: PICC: number analyzed (Participants) | 19 | 1
  Cycle 8 Day 1: Q1d: PICC | 47.4 | 100
  Cycle 8 Day 1: Q1d: Port-a-Cath: number analyzed (Participants) | 19 | 1
  Cycle 8 Day 1: Q1d: Port-a-Cath | 31.6 | 0
  Cycle 8 Day 1: Q1d: Tunneled Central Venous Catheter: number analyzed (Participants) | 19 | 1
  Cycle 8 Day 1: Q1d: Tunneled Central Venous Catheter | 10.5 | 0
  Cycle 8 Day 1: Q1e: Within 7 Days Prior Today: number analyzed (Participants) | 15 | 14
  Cycle 8 Day 1: Q1e: Within 7 Days Prior Today | 20.0 | 14.3
  Cycle 8 Day 1: Q1e: > 7 < 14 Days Prior Today: number analyzed (Participants) | 15 | 14
  Cycle 8 Day 1: Q1e: > 7 < 14 Days Prior Today | 13.3 | 28.6
  Cycle 8 Day 1: Q1e: > 14 < 30 Days Prior Today: number analyzed (Participants) | 15 | 14
  Cycle 8 Day 1: Q1e: > 14 < 30 Days Prior Today | 20.0 | 0
  Cycle 8 Day 1: Q1e: Other: number analyzed (Participants) | 15 | 14
  Cycle 8 Day 1: Q1e: Other | 46.7 | 57.1

6. Secondary Outcome: Neoadjuvant Phase: Duration of Treatment Administration According to HCPs' Responses to Questions 1c (Sub-part), 1f, and 1g of the HCPQ - Administering Treatment
Description: HCP was defined as any personnel involved in the drug preparation and/or drug administration processes. HCPs who have had experience with administration of P+H IV and/or PH FDC SC completed the following Questions of the HCPQ: Q1c: If new IV access was needed for this cycle of treatment, how long (in minutes) this took to set up? Q1f: How long (in minutes) did it take to administer the treatment (P+H IV or PH FDC SC)? Q1g: How long (in minutes) was the participant in the Treatment Area in total? Percentages have been rounded off.
Time Frame: Day 1 of Cycles 1-8 (Cycle length = 21 days)
Population: Overall number analyzed is the number of HCPs who answered Q1c, Q1f and Q1g of the HCPQ. Number analyzed is the number of HCPs who answered Q1c, Q1f and Q1g of the HCPQ at the specified time point.
Measure: Median (Full Range); unit: minutes
Arm/Group | Arm A, Neoadjuvant Phase: P+H IV | Arm B, Neoadjuvant Phase: PH FDC SC
Number analyzed (Participants) | 112 | 212
minutes
  Cycle 1 Day 1: Q1c: number analyzed (Participants) | 46 | 8
  Cycle 1 Day 1: Q1c | 5.0 [1 to 150] | 5.0 [1 to 308]
  Cycle 1 Day 1: Q1f: number analyzed (Participants) | 61 | 121
  Cycle 1 Day 1: Q1f | 180.0 [60 to 390] | 8.0 [5 to 30]
  Cycle 1 Day 1: Q1g: number analyzed (Participants) | 63 | 121
  Cycle 1 Day 1: Q1g | 420.0 [120 to 520] | 180.0 [8 to 424]
  Cycle 2 Day 1: Q1c: number analyzed (Participants) | 46 | 3
  Cycle 2 Day 1: Q1c | 5.0 [1 to 18] | 5.0 [2 to 6]
  Cycle 2 Day 1: Q1f: number analyzed (Participants) | 58 | 118
  Cycle 2 Day 1: Q1f | 82.5 [5 to 360] | 5.0 [5 to 190]
  Cycle 2 Day 1: Q1g: number analyzed (Participants) | 62 | 118
  Cycle 2 Day 1: Q1g | 300.0 [90 to 503] | 180.0 [5 to 330]
  Cycle 3 Day 1: Q1c: number analyzed (Participants) | 43 | 5
  Cycle 3 Day 1: Q1c | 5.0 [1 to 20] | 10.0 [5 to 10]
  Cycle 3 Day 1: Q1f: number analyzed (Participants) | 59 | 111
  Cycle 3 Day 1: Q1f | 90.0 [5 to 360] | 5.0 [3 to 159]
  Cycle 3 Day 1: Q1g: number analyzed (Participants) | 61 | 111
  Cycle 3 Day 1: Q1g | 280.0 [90 to 500] | 180.0 [6 to 480]
  Cycle 4 Day 1: Q1c: number analyzed (Participants) | 40 | 4
  Cycle 4 Day 1: Q1c | 5.0 [2 to 20] | 6.5 [5 to 10]
  Cycle 4 Day 1: Q1f: number analyzed (Participants) | 57 | 112
  Cycle 4 Day 1: Q1f | 90.0 [14 to 365] | 5.0 [3 to 15]
  Cycle 4 Day 1: Q1g: number analyzed (Participants) | 61 | 113
  Cycle 4 Day 1: Q1g | 270.0 [30 to 560] | 170.0 [6 to 480]
  Cycle 5 Day 1: Q1c: number analyzed (Participants) | 71 | 5
  Cycle 5 Day 1: Q1c | 5.0 [1 to 150] | 5.0 [1 to 10]
  Cycle 5 Day 1: Q1f: number analyzed (Participants) | 108 | 210
  Cycle 5 Day 1: Q1f | 145.0 [8 to 360] | 8.0 [4 to 250]
  Cycle 5 Day 1: Q1g | 294.0 [30 to 552] | 150.0 [5 to 420]
  Cycle 6 Day 1: Q1c: number analyzed (Participants) | 74 | 6
  Cycle 6 Day 1: Q1c | 5.0 [1 to 25] | 5.0 [2 to 5]
  Cycle 6 Day 1: Q1f: number analyzed (Participants) | 108 | 204
  Cycle 6 Day 1: Q1f | 90.0 [8 to 360] | 5.0 [4 to 80]
  Cycle 6 Day 1: Q1g: number analyzed (Participants) | 109 | 203
  Cycle 6 Day 1: Q1g | 260.0 [35 to 510] | 150.0 [5 to 370]
  Cycle 7 Day 1: Q1c: number analyzed (Participants) | 41 | 1
  Cycle 7 Day 1: Q1c | 5.0 [1 to 30] | 3.0 [3 to 3]
  Cycle 7 Day 1: Q1f: number analyzed (Participants) | 57 | 110
  Cycle 7 Day 1: Q1f | 90.0 [8 to 210] | 5.0 [4 to 75]
  Cycle 7 Day 1: Q1g: number analyzed (Participants) | 57 | 111
  Cycle 7 Day 1: Q1g | 190.0 [40 to 480] | 115.0 [5 to 360]
  Cycle 8 Day 1: Q1c: number analyzed (Participants) | 38 | 5
  Cycle 8 Day 1: Q1c | 5.0 [1 to 20] | 5.0 [4 to 8]
  Cycle 8 Day 1: Q1f: number analyzed (Participants) | 57 | 106
  Cycle 8 Day 1: Q1f | 90.0 [5 to 180] | 5.0 [3 to 25]
  Cycle 8 Day 1: Q1g: number analyzed (Participants) | 57 | 106
  Cycle 8 Day 1: Q1g | 180.0 [60 to 535] | 120.0 [6 to 345]

7. Secondary Outcome: Neoadjuvant Phase: Percentage of HCPs by Their Response to Question 2 (2a to 2e) of the HCPQ - Administering Treatment
Description: HCP was defined as any personnel involved in the drug preparation &/or drug administration processes. HCPs who have had experience with administration of P+H IV &/or PH FDC SC completed Q2 (2a-2e) of the HCPQ: In your opinion, if all P+H IV infusions were switched to PH FDC SC injections, please indicate how strongly you agree/disagree with each of the following statements. 2a: Participants may be moved out of the Treatment Area (for infusion treatment) to receive PH FDC SC injections. 2b: PH FDC SC's SC route of administration allows for more flexible treatment scheduling. 2c: Frees up infusion chairs for participants whose treatments can only be given IV. 2d: Waiting list for any P+H IV treatment at the Treatment Area is reduced. 2e: Staff's work burden is reduced, enhancing work performance. The 6 available options were: Strongly Disagree, Disagree, Neutral, Agree, Strongly Agree and Not applicable. Percentages were rounded off.
Time Frame: Up to Cycle 8 (Cycle length = 21 days)
Population: Overall number analyzed is the number of HCPs who answered any sub part Q2 (2a to 2e) of the HCPQ. Number analyzed is the number of HCPs who answered each sub-question of Q2 (2a to 2e) of the HCPQ.
Measure: Number; unit: percentage of HCPs
Arm/Group | Arm A, Neoadjuvant Phase: P+H IV | Arm B, Neoadjuvant Phase: PH FDC SC
Number analyzed (Participants) | 98 | 166
percentage of HCPs
  Q2a: Strongly Disagree: number analyzed (Participants) | 97 | 164
  Q2a: Strongly Disagree | 1.0 | 3.0
  Q2a: Disagree: number analyzed (Participants) | 97 | 164
  Q2a: Disagree | 8.2 | 13.4
  Q2a: Neutral: number analyzed (Participants) | 97 | 164
  Q2a: Neutral | 14.4 | 13.4
  Q2a: Agree: number analyzed (Participants) | 97 | 164
  Q2a: Agree | 36.1 | 28.7
  Q2a: Strongly Agree: number analyzed (Participants) | 97 | 164
  Q2a: Strongly Agree | 32.0 | 33.5
  Q2a: Not Applicable: number analyzed (Participants) | 97 | 164
  Q2a: Not Applicable | 8.2 | 7.9
  Q2b: Strongly Disagree | 0 | 2.4
  Q2b: Disagree | 9.2 | 6.0
  Q2b: Neutral | 12.2 | 13.9
  Q2b: Agree | 37.8 | 34.3
  Q2b: Strongly Agree | 33.7 | 35.5
  Q2b: Not Applicable | 7.1 | 7.8
  Q2c: Strongly Disagree | 1.0 | 3.0
  Q2c: Disagree | 9.2 | 6.0
  Q2c: Neutral | 10.2 | 10.8
  Q2c: Agree | 32.7 | 35.5
  Q2c: Strongly Agree | 39.8 | 37.3
  Q2c: Not Applicable | 7.1 | 7.2
  Q2d: Strongly Disagree | 0 | 1.8
  Q2d: Disagree | 8.2 | 6.0
  Q2d: Neutral | 15.3 | 15.7
  Q2d: Agree | 34.7 | 37.3
  Q2d: Strongly Agree | 35.7 | 31.9
  Q2d: Not Applicable | 6.1 | 7.2
  Q2e: Strongly Disagree: number analyzed (Participants) | 98 | 165
  Q2e: Strongly Disagree | 0 | 3.6
  Q2e: Disagree: number analyzed (Participants) | 98 | 165
  Q2e: Disagree | 5.1 | 3.6
  Q2e: Neutral: number analyzed (Participants) | 98 | 165
  Q2e: Neutral | 27.6 | 25.5
  Q2e: Agree: number analyzed (Participants) | 98 | 165
  Q2e: Agree | 26.5 | 27.3
  Q2e: Strongly Agree: number analyzed (Participants) | 98 | 165
  Q2e: Strongly Agree | 34.7 | 32.7
  Q2e: Not Applicable: number analyzed (Participants) | 98 | 165
  Q2e: Not Applicable | 6.1 | 7.3

8. Secondary Outcome: Neoadjuvant Phase: Percentage of HCPs by Their Responses to Question 2 (2f to 2j) of the HCPQ - Administering Treatment
Description: HCP was defined as any personnel involved in the drug preparation &/or drug administration processes. HCPs who have had experience with administration of P+H IV &/or PH FDC SC completed Question 2 (2f to 2j) of the HCPQ: In your opinion, if all P+H IV infusions were switched to PH FDC SC injections, please indicate how strongly you agree/disagree with each of the following statements. 2f: More interaction time between HCPs and participants. 2g: Staff have more time for further professional education/development. 2h: Staff has more time for administrative tasks. 2i: Participants on PH FDC SC spend less time in the Treatment Area. 2j: Participants prefer PH FDC SC to P+H IV. The 6 available options were: Strongly Disagree, Disagree, Neutral, Agree, Strongly Agree and Not applicable. Percentages were rounded off.
Time Frame: Up to Cycle 8 (Cycle length = 21 days)
Population: Overall number analyzed is the number of HCPs who answered any sub part of Q2 (2f to 2j) of the HCPQ. Number analyzed is the number of HCPs who answered each sub-question of Q2 (2f to 2j) of the HCPQ.
Measure: Number; unit: percentage of HCPs
Arm/Group | Arm A, Neoadjuvant Phase: P+H IV | Arm B, Neoadjuvant Phase: PH FDC SC
Number analyzed (Participants) | 98 | 166
percentage of HCPs
  Q2f: Strongly Disagree | 0 | 2.4
  Q2f: Disagree | 8.2 | 4.2
  Q2f: Neutral | 20.4 | 34.3
  Q2f: Agree | 33.7 | 22.3
  Q2f: Strongly Agree | 31.6 | 28.9
  Q2f: Not Applicable | 6.1 | 7.8
  Q2g: Strongly Disagree | 2.0 | 2.4
  Q2g: Disagree | 5.1 | 4.8
  Q2g: Neutral | 25.5 | 36.7
  Q2g: Agree | 31.6 | 22.9
  Q2g: Strongly Agree | 29.6 | 25.3
  Q2g: Not Applicable | 6.1 | 7.8
  Q2h: Strongly Disagree | 0 | 1.2
  Q2h: Disagree | 6.1 | 3.6
  Q2h: Neutral | 23.5 | 31.9
  Q2h: Agree | 30.6 | 25.9
  Q2h: Strongly Agree | 33.7 | 28.9
  Q2h: Not Applicable | 6.1 | 8.4
  Q2i: Strongly Disagree: number analyzed (Participants) | 97 | 166
  Q2i: Strongly Disagree | 1.0 | 1.8
  Q2i: Disagree: number analyzed (Participants) | 97 | 166
  Q2i: Disagree | 0 | 1.8
  Q2i: Neutral: number analyzed (Participants) | 97 | 166
  Q2i: Neutral | 4.1 | 3.0
  Q2i: Agree: number analyzed (Participants) | 97 | 166
  Q2i: Agree | 26.8 | 31.9
  Q2i: Strongly Agree: number analyzed (Participants) | 97 | 166
  Q2i: Strongly Agree | 61.9 | 53.0
  Q2i: Not Applicable: number analyzed (Participants) | 97 | 166
  Q2i: Not Applicable | 6.2 | 8.4
  Q2j: Strongly Disagree: number analyzed (Participants) | 97 | 166
  Q2j: Strongly Disagree | 1.0 | 0.6
  Q2j: Disagree: number analyzed (Participants) | 97 | 166
  Q2j: Disagree | 1.0 | 1.8
  Q2j: Neutral: number analyzed (Participants) | 97 | 166
  Q2j: Neutral | 20.6 | 21.7
  Q2j: Agree: number analyzed (Participants) | 97 | 166
  Q2j: Agree | 35.1 | 31.3
  Q2j: Strongly Agree: number analyzed (Participants) | 97 | 166
  Q2j: Strongly Agree | 35.1 | 32.5
  Q2j: Not Applicable: number analyzed (Participants) | 97 | 166
  Q2j: Not Applicable | 7.2 | 12.0

9. Secondary Outcome: Neoadjuvant Phase: Percentage of HCPs by Their Responses to Question 3 to 11 of the HCPQ - Administering Treatment
Description: HCPs who have had experience with administration of P+H IV &/or PH FDC SC completed Questions 3 to 11 of the HCPQ: Q3: Which was more convenient for the participant? Q4: Which was better for optimising participant care at your institution? Q5: Which required less time to administer (excluding observation period)? Q6: Which required less use of institutional resources (e.g., staff time, facility costs, equipment use)? Q7: Which required less time to administer all the treatment (including IV chemotherapy)? Q8: Which allowed for attending to more participants because of time savings from the mode of administration of pertuzumab and trastuzumab? Q9: During the NP you had to administer IV chemotherapy through participant's IV access. You prefer to accompany IV chemotherapy with? Q10: Which was preferred by participants? Q11: How frequently would you recommend PH FDC SC administration to your participants in the future? Percentages were rounded off.
Time Frame: Up to Cycle 8 (Cycle length = 21 days)
Population: Overall number analyzed is the number of HCPs who answered any of the questions from Q3 to Q11 of the HCPQ. Number analyzed is the number of HCPs who answered each specific question (Q3 to Q11) of the HCPQ.
Measure: Number; unit: percentage of HCPs
Arm/Group | Arm A, Neoadjuvant Phase: P+H IV | Arm B, Neoadjuvant Phase: PH FDC SC
Number analyzed (Participants) | 98 | 166
percentage of HCPs
  Q3: P+H IV: number analyzed (Participants) | 88 | 161
  Q3: P+H IV | 8.0 | 1.2
  Q3: PH FDC SC: number analyzed (Participants) | 88 | 161
  Q3: PH FDC SC | 68.2 | 83.9
  Q3: No Difference: number analyzed (Participants) | 88 | 161
  Q3: No Difference | 13.6 | 8.7
  Q3: Unsure: number analyzed (Participants) | 88 | 161
  Q3: Unsure | 10.2 | 6.2
  Q4: P+H IV: number analyzed (Participants) | 88 | 162
  Q4: P+H IV | 5.7 | 1.9
  Q4: PH FDC SC: number analyzed (Participants) | 88 | 162
  Q4: PH FDC SC | 69.3 | 82.1
  Q4: No Difference: number analyzed (Participants) | 88 | 162
  Q4: No Difference | 22.7 | 13.0
  Q4: Unsure: number analyzed (Participants) | 88 | 162
  Q4: Unsure | 2.3 | 3.1
  Q5: P+H IV: number analyzed (Participants) | 88 | 162
  Q5: P+H IV | 0 | 0.6
  Q5: PH FDC SC: number analyzed (Participants) | 88 | 162
  Q5: PH FDC SC | 92.0 | 97.5
  Q5: No Difference: number analyzed (Participants) | 88 | 162
  Q5: No Difference | 8.0 | 1.9
  Q5: Unsure: number analyzed (Participants) | 88 | 162
  Q5: Unsure | 0 | 0
  Q6: P+H IV: number analyzed (Participants) | 88 | 162
  Q6: P+H IV | 0 | 0.6
  Q6: PH FDC SC: number analyzed (Participants) | 88 | 162
  Q6: PH FDC SC | 83.0 | 88.9
  Q6: No Difference: number analyzed (Participants) | 88 | 162
  Q6: No Difference | 17.0 | 10.5
  Q6: Unsure: number analyzed (Participants) | 88 | 162
  Q6: Unsure | 0 | 0
  Q7: P+H IV: number analyzed (Participants) | 88 | 162
  Q7: P+H IV | 1.1 | 0
  Q7: PH FDC SC: number analyzed (Participants) | 88 | 162
  Q7: PH FDC SC | 96.6 | 98.1
  Q7: No Difference: number analyzed (Participants) | 88 | 162
  Q7: No Difference | 2.3 | 1.9
  Q7: Unsure: number analyzed (Participants) | 88 | 162
  Q7: Unsure | 0 | 0
  Q8: P+H IV: number analyzed (Participants) | 87 | 162
  Q8: P+H IV | 0 | 0.6
  Q8: PH FDC SC: number analyzed (Participants) | 87 | 162
  Q8: PH FDC SC | 73.6 | 82.7
  Q8: No Difference: number analyzed (Participants) | 87 | 162
  Q8: No Difference | 26.4 | 16.7
  Q8: Unsure: number analyzed (Participants) | 87 | 162
  Q8: Unsure | 0 | 0
  Q9: P+H IV: number analyzed (Participants) | 87 | 161
  Q9: P+H IV | 12.6 | 8.7
  Q9: PH FDC SC: number analyzed (Participants) | 87 | 161
  Q9: PH FDC SC | 73.6 | 73.9
  Q9: No Difference: number analyzed (Participants) | 87 | 161
  Q9: No Difference | 13.8 | 17.4
  Q9: Unsure: number analyzed (Participants) | 87 | 161
  Q9: Unsure | 0 | 0
  Q10: P+H IV: number analyzed (Participants) | 89 | 162
  Q10: P+H IV | 7.9 | 1.2
  Q10: PH FDC SC: number analyzed (Participants) | 89 | 162
  Q10: PH FDC SC | 66.3 | 73.5
  Q10: No Difference: number analyzed (Participants) | 89 | 162
  Q10: No Difference | 10.1 | 7.4
  Q10: Unsure: number analyzed (Participants) | 89 | 162
  Q10: Unsure | 15.7 | 17.9
  Q11: Always: number analyzed (Participants) | 89 | 158
  Q11: Always | 75.3 | 79.1
  Q11: Sometimes: number analyzed (Participants) | 89 | 158
  Q11: Sometimes | 24.7 | 19.0
  Q11: Never: number analyzed (Participants) | 89 | 158
  Q11: Never | 0 | 1.9

10. Secondary Outcome: Percentage of Participants Who Achieved pCR Post-surgery
Description: pCR was defined as the absence of residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy (i.e., ypT0/Tis ypN0), according to the current American Joint Committee on Cancer (AJCC) staging system classification. Percentages were rounded off.
Time Frame: Up to approximately 7.8 months
Population: FASab included all randomized participants, regardless of whether they received treatment. Overall number analyzed is the number of participants with data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A, Neoadjuvant Phase: P+H IV | Arm B, Neoadjuvant Phase: PH FDC SC
Number analyzed (Participants) | 113 | 207
percentage of participants | 60.2 | 60.9

11. Secondary Outcome: Neoadjuvant Phase: Change From Baseline in Health-related Quality of Life (HRQoL) Assessed by European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQ C30) Scores
Description: EORTC QLQ-C30=cancer-specific instrument consisting of 30 questions that evaluated 5 aspects of participant functioning (physical, emotional, role, cognitive & social), 3 symptom scales (fatigue, nausea & vomiting & pain), global health status/quality of life (GHS/QoL) & 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea & financial difficulties). Functioning & symptom items used a 4-point scale, scores ranging from 1=Not at all to 4=Very much. GHS/QoL questions used a 7-point scale, scores ranging from 1=Very poor to 7=Excellent. All EORTC scales & single-item measures were linearly transformed to a score range of 0-100. High score for functional/GHS scale=high/healthy level of functioning/better HRQoL & high score for symptom scale=high level of symptom severity. A positive change from baseline=improvement & negative change=worsening in QoL & functioning scales. A positive change from baseline=deterioration & negative change=improvement in symptom scales.
Time Frame: Baseline, Day 1 of Cycles 6 and 8 (Cycle length = 21 days)
Population: FASab included all randomized participants, regardless of whether they received treatment. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A, Neoadjuvant Phase: P+H IV | Arm B, Neoadjuvant Phase: PH FDC SC
Number analyzed (Participants) | 115 | 223
score on a scale
  Baseline - GHS/QoL | 79.86 (18.40) | 75.97 (20.92)
  Change at Cycle 6 Day 1 - GHS/QoL: number analyzed (Participants) | 61 | 107
  Change at Cycle 6 Day 1 - GHS/QoL | -9.43 (21.27) | -7.40 (24.64)
  Change at Cycle 8 Day 1 - GHS/QoL: number analyzed (Participants) | 52 | 95
  Change at Cycle 8 Day 1 - GHS/QoL | -10.42 (19.73) | -11.75 (26.78)
  Baseline - Physical functioning (PF) | 91.65 (11.84) | 91.84 (12.45)
  Change at Cycle 6 Day 1 - PF: number analyzed (Participants) | 61 | 107
  Change at Cycle 6 Day 1 - PF | -12.65 (16.18) | -16.01 (18.56)
  Change at Cycle 8 Day 1 - PF: number analyzed (Participants) | 52 | 95
  Change at Cycle 8 Day 1 - PF | -16.03 (19.28) | -13.00 (16.25)
  Baseline - Role Functioning (RF) | 91.88 (15.82) | 91.48 (19.11)
  Change at Cycle 6 Day 1 - RF: number analyzed (Participants) | 61 | 107
  Change at Cycle 6 Day 1 - RF | -15.85 (28.78) | -21.18 (29.46)
  Change at Cycle 8 Day 1 - RF: number analyzed (Participants) | 52 | 95
  Change at Cycle 8 Day 1 - RF | -19.87 (27.62) | -14.91 (27.98)
  Baseline - Emotional Functioning (EF) | 73.41 (22.13) | 71.45 (22.54)
  Change at Cycle 6 Day 1 - EF: number analyzed (Participants) | 61 | 107
  Change at Cycle 6 Day 1 - EF | -5.87 (26.06) | 1.01 (25.20)
  Change at Cycle 8 Day 1 - EF: number analyzed (Participants) | 52 | 95
  Change at Cycle 8 Day 1 - EF | 5.29 (24.09) | 5.85 (25.01)
  Baseline - Cognitive functioning (CF) | 88.41 (19.01) | 88.19 (17.62)
  Change at Cycle 6 Day 1 - CF: number analyzed (Participants) | 61 | 107
  Change at Cycle 6 Day 1 - CF | -12.02 (22.39) | -10.28 (23.53)
  Change at Cycle 8 Day 1 - CF: number analyzed (Participants) | 52 | 95
  Change at Cycle 8 Day 1 - CF | -9.62 (25.21) | -4.74 (18.78)
  Baseline - Social Functioning (SF) | 86.67 (22.96) | 84.30 (24.56)
  Change at Cycle 6 Day 1 - SF: number analyzed (Participants) | 61 | 107
  Change at Cycle 6 Day 1 - SF | -18.03 (30.01) | -15.26 (32.55)
  Change at Cycle 8 Day 1 - SF: number analyzed (Participants) | 52 | 95
  Change at Cycle 8 Day 1 - SF | -14.42 (27.82) | -7.54 (25.59)
  Baseline - Fatigue | 15.85 (20.29) | 16.44 (17.74)
  Change at Cycle 6 Day 1 - Fatigue: number analyzed (Participants) | 61 | 107
  Change at Cycle 6 Day 1 - Fatigue | 24.04 (26.23) | 27.21 (25.91)
  Change at Cycle 8 Day 1 - Fatigue: number analyzed (Participants) | 52 | 95
  Change at Cycle 8 Day 1 - Fatigue | 23.29 (24.33) | 20.23 (24.31)
  Baseline - Nausea & Vomiting | 4.06 (11.60) | 3.36 (10.25)
  Change at Cycle 6 Day 1 - Nausea & Vomiting: number analyzed (Participants) | 61 | 107
  Change at Cycle 6 Day 1 - Nausea & Vomiting | 19.95 (24.69) | 14.80 (22.82)
  Change at Cycle 8 Day 1 - Nausea & Vomiting: number analyzed (Participants) | 52 | 95
  Change at Cycle 8 Day 1 - Nausea & Vomiting | 3.21 (20.88) | 4.74 (17.64)
  Baseline - Pain | 12.17 (18.25) | 14.13 (19.14)
  Change at Cycle 6 Day 1 - Pain: number analyzed (Participants) | 61 | 107
  Change at Cycle 6 Day 1 - Pain | 14.21 (27.53) | 7.79 (25.83)
  Change at Cycle 8 Day 1 - Pain: number analyzed (Participants) | 52 | 95
  Change at Cycle 8 Day 1 - Pain | 11.86 (29.21) | 8.07 (21.59)
  Baseline - Dyspnoea | 4.35 (14.32) | 6.28 (16.45)
  Change at Cycle 6 Day 1 - Dyspnoea: number analyzed (Participants) | 61 | 107
  Change at Cycle 6 Day 1 - Dyspnoea | 8.74 (23.49) | 12.46 (24.88)
  Change at Cycle 8 Day 1 - Dyspnoea: number analyzed (Participants) | 52 | 95
  Change at Cycle 8 Day 1 - Dyspnoea | 13.46 (28.97) | 6.67 (23.11)
  Baseline - Insomnia | 25.22 (30.14) | 24.51 (28.07)
  Change at Cycle 6 Day 1 - Insomnia: number analyzed (Participants) | 61 | 107
  Change at Cycle 6 Day 1 - Insomnia | 4.37 (32.48) | 3.12 (35.33)
  Change at Cycle 8 Day 1 - Insomnia: number analyzed (Participants) | 52 | 95
  Change at Cycle 8 Day 1 - Insomnia | 8.97 (40.75) | 9.12 (33.84)
  Baseline - Appetite Loss | 8.41 (20.16) | 9.72 (20.51)
  Change at Cycle 6 Day 1 - Appetite Loss: number analyzed (Participants) | 61 | 107
  Change at Cycle 6 Day 1 - Appetite Loss | 21.31 (32.22) | 23.99 (33.89)
  Change at Cycle 8 Day 1 - Appetite Loss: number analyzed (Participants) | 52 | 95
  Change at Cycle 8 Day 1 - Appetite Loss | 16.03 (33.97) | 15.09 (35.65)
  Baseline - Constipation | 9.57 (21.07) | 9.87 (20.56)
  Change at Cycle 6 Day 1 - Constipation: number analyzed (Participants) | 61 | 107
  Change at Cycle 6 Day 1 - Constipation | 7.65 (29.44) | 5.61 (25.69)
  Change at Cycle 8 Day 1 - Constipation: number analyzed (Participants) | 51 | 95
  Change at Cycle 8 Day 1 - Constipation | 2.61 (21.95) | 3.86 (24.73)
  Baseline - Diarrhoea | 3.77 (13.07) | 4.93 (14.86)
  Change at Cycle 6 Day 1 - Diarrhoea: number analyzed (Participants) | 61 | 107
  Change at Cycle 6 Day 1 - Diarrhoea | 25.68 (33.55) | 28.04 (34.31)
  Change at Cycle 8 Day 1 - Diarrhoea: number analyzed (Participants) | 52 | 95
  Change at Cycle 8 Day 1 - Diarrhoea | 32.05 (26.37) | 27.37 (33.68)
  Baseline - Financial Difficulties | 26.09 (34.14) | 23.17 (32.67)
  Change at Cycle 6 Day 1 - Financial Difficulties: number analyzed (Participants) | 61 | 107
  Change at Cycle 6 Day 1 - Financial Difficulties | 6.01 (41.95) | 7.79 (35.93)
  Change at Cycle 8 Day 1 - Financial Difficulties: number analyzed (Participants) | 52 | 95
  Change at Cycle 8 Day 1 - Financial Difficulties | 6.41 (28.80) | -1.40 (33.66)

12. Secondary Outcome: Adjuvant Phase: Change From Baseline in HRQoL Assessed by EORTC QLQ C30 Scores
Description: EORTC QLQ-C30=cancer-specific instrument consisting of 30 questions that evaluated 5 aspects of participant functioning (physical, emotional, role, cognitive & social), 3 symptom scales (fatigue, nausea & vomiting & pain), GHS/QoL & 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea & financial difficulties). Functioning & symptom items used a 4-point scale, scores ranging from 1=Not at all to 4=Very much. GHS/QoL questions used a 7-point scale, scores ranging from 1=Very poor to 7=Excellent. All EORTC scales & single-item measures were linearly transformed to a score range of 0-100. High score for functional/GHS scale=high/healthy level of functioning/better HRQoL & high score for symptom scale=high level of symptom severity. A positive change from baseline=improvement & negative change=worsening in QoL & functioning scales. A positive change from baseline=deterioration & negative change=improvement in symptom scales.
Time Frame: Baseline (Cycle 1) of Run-in Period; Day 1 of Cycles 1, 3, and 6 in the Cross-over Period (Cycle length = 21 days)
Population: mITTcross population included all randomized participants assigned into the cross-over period who received at least one dose of PH FDC SC, completed Question 1 of the PPQ and completed radiotherapy before entering the cross-over period. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm C, Adjuvant Cross-over Phase: PH FDC SC in Hospital, Then at Home | Arm D, Adjuvant Cross-Over Phase: PH FDC SC at Home, Then in Hospital
Number analyzed (Participants) | 98 | 96
score on a scale
  Baseline - GHS/QoL: number analyzed (Participants) | 97 | 96
  Baseline - GHS/QoL | 76.98 (17.09) | 71.79 (18.63)
  Change at Cycle 1 Day 1- GHS/QoL: number analyzed (Participants) | 89 | 91
  Change at Cycle 1 Day 1- GHS/QoL | 0.66 (13.72) | 0.09 (18.57)
  Change at Cycle 3 Day 1 - GHS/QoL: number analyzed (Participants) | 88 | 89
  Change at Cycle 3 Day 1 - GHS/QoL | 2.08 (14.53) | 5.15 (20.59)
  Change at Cycle 6 Day 1 - GHS/QoL: number analyzed (Participants) | 88 | 84
  Change at Cycle 6 Day 1 - GHS/QoL | -0.57 (16.61) | 2.48 (19.99)
  Baseline - Physical Functioning (PF): number analyzed (Participants) | 97 | 96
  Baseline - Physical Functioning (PF) | 82.61 (15.89) | 80.35 (16.20)
  Change at Cycle 1 Day 1 - PF: number analyzed (Participants) | 88 | 91
  Change at Cycle 1 Day 1 - PF | 2.50 (13.19) | 1.83 (14.44)
  Change at Cycle 3 Day 1 - PF: number analyzed (Participants) | 88 | 91
  Change at Cycle 3 Day 1 - PF | 2.50 (13.65) | 5.99 (14.18)
  Change at Cycle 6 Day 1 - PF: number analyzed (Participants) | 88 | 84
  Change at Cycle 6 Day 1 - PF | 4.13 (16.97) | 2.46 (14.99)
  Baseline - Role Functioning (RF): number analyzed (Participants) | 97 | 96
  Baseline - Role Functioning (RF) | 78.35 (21.40) | 66.67 (29.72)
  Change at Cycle 1 Day 1 - RF: number analyzed (Participants) | 88 | 91
  Change at Cycle 1 Day 1 - RF | 4.92 (21.61) | 10.62 (27.84)
  Change at Cycle 3 Day 1 - RF: number analyzed (Participants) | 88 | 89
  Change at Cycle 3 Day 1 - RF | 6.25 (23.61) | 17.23 (31.33)
  Change at Cycle 6 Day 1 - RF: number analyzed (Participants) | 88 | 84
  Change at Cycle 6 Day 1 - RF | 9.66 (23.53) | 16.07 (31.73)
  Baseline - Emotional Functioning (EF): number analyzed (Participants) | 97 | 96
  Baseline - Emotional Functioning (EF) | 82.22 (19.31) | 76.65 (22.61)
  Change at Cycle 1 Day 1 - EF: number analyzed (Participants) | 89 | 91
  Change at Cycle 1 Day 1 - EF | -1.22 (18.44) | 0.34 (23.55)
  Change at Cycle 3 Day 1 - EF: number analyzed (Participants) | 88 | 89
  Change at Cycle 3 Day 1 - EF | 2.27 (16.75) | 3.46 (18.84)
  Change at Cycle 6 Day 1 - EF: number analyzed (Participants) | 88 | 84
  Change at Cycle 6 Day 1 - EF | -0.95 (21.86) | 0.60 (19.86)
  Baseline - Cognitive Functioning (CF): number analyzed (Participants) | 97 | 96
  Baseline - Cognitive Functioning (CF) | 84.54 (21.14) | 79.51 (24.24)
  Change at Cycle 1 Day 1 - CF: number analyzed (Participants) | 89 | 91
  Change at Cycle 1 Day 1 - CF | -3.37 (21.05) | 0.00 (22.50)
  Change at Cycle 3 Day 1 - CF: number analyzed (Participants) | 88 | 89
  Change at Cycle 3 Day 1 - CF | -2.08 (21.11) | 1.12 (21.14)
  Change at Cycle 6 Day 1 - CF: number analyzed (Participants) | 88 | 84
  Change at Cycle 6 Day 1 - CF | -2.65 (22.30) | 0.00 (24.54)
  Baseline - Social Functioning (SF): number analyzed (Participants) | 97 | 96
  Baseline - Social Functioning (SF) | 80.58 (22.65) | 70.49 (25.87)
  Change at Cycle 1 Day 1 - SF: number analyzed (Participants) | 89 | 91
  Change at Cycle 1 Day 1 - SF | 1.69 (22.34) | 6.59 (27.76)
  Change at Cycle 3 Day 1 - SF: number analyzed (Participants) | 88 | 89
  Change at Cycle 3 Day 1 - SF | 1.70 (20.69) | 9.74 (25.23)
  Change at Cycle 6 Day 1 - SF: number analyzed (Participants) | 88 | 84
  Change at Cycle 6 Day 1 - SF | 0.95 (21.64) | 9.92 (25.89)
  Baseline - Fatigue: number analyzed (Participants) | 97 | 96
  Baseline - Fatigue | 26.92 (21.92) | 31.83 (23.56)
  Change at Cycle 1 Day 1 - Fatigue: number analyzed (Participants) | 89 | 91
  Change at Cycle 1 Day 1 - Fatigue | -3.62 (17.55) | -0.61 (24.31)
  Change at Cycle 3 Day 1 - Fatigue: number analyzed (Participants) | 88 | 89
  Change at Cycle 3 Day 1 - Fatigue | -3.66 (18.66) | -7.99 (21.65)
  Change at Cycle 6 Day 1 - Fatigue: number analyzed (Participants) | 88 | 84
  Change at Cycle 6 Day 1 - Fatigue | -4.42 (24.09) | -4.37 (23.84)
  Baseline - Nausea & Vomiting: number analyzed (Participants) | 97 | 96
  Baseline - Nausea & Vomiting | 4.64 (10.96) | 5.38 (11.47)
  Change at Cycle 1 Day 1 - Nausea & Vomiting: number analyzed (Participants) | 88 | 91
  Change at Cycle 1 Day 1 - Nausea & Vomiting | -0.95 (11.95) | 1.83 (14.79)
  Change at Cycle 3 Day 1 - Nausea & Vomiting: number analyzed (Participants) | 88 | 89
  Change at Cycle 3 Day 1 - Nausea & Vomiting | -0.57 (11.43) | -1.31 (10.43)
  Change at Cycle 6 Day 1 - Nausea & Vomiting: number analyzed (Participants) | 88 | 84
  Change at Cycle 6 Day 1 - Nausea & Vomiting | -0.95 (12.21) | 0.99 (12.77)
  Baseline - Pain: number analyzed (Participants) | 97 | 96
  Baseline - Pain | 22.51 (20.84) | 28.82 (26.10)
  Change at Cycle 1 Day 1 - Pain: number analyzed (Participants) | 88 | 91
  Change at Cycle 1 Day 1 - Pain | -5.30 (21.82) | -7.14 (23.46)
  Change at Cycle 3 Day 1 - Pain: number analyzed (Participants) | 89 | 89
  Change at Cycle 3 Day 1 - Pain | -6.37 (20.18) | -9.74 (25.97)
  Change at Cycle 6 Day 1 - Pain: number analyzed (Participants) | 88 | 84
  Change at Cycle 6 Day 1 - Pain | -6.06 (23.59) | -8.73 (27.19)
  Baseline - Dyspnoea: number analyzed (Participants) | 97 | 96
  Baseline - Dyspnoea | 7.56 (17.68) | 8.68 (17.60)
  Change at Cycle 1 Day 1 - Dyspnoea: number analyzed (Participants) | 88 | 91
  Change at Cycle 1 Day 1 - Dyspnoea | 1.89 (20.44) | 0.73 (21.65)
  Change at Cycle 3 Day 1 - Dyspnoea: number analyzed (Participants) | 88 | 89
  Change at Cycle 3 Day 1 - Dyspnoea | 0.00 (20.84) | 0.75 (21.89)
  Change at Cycle 6 Day 1 - Dyspnoea: number analyzed (Participants) | 88 | 84
  Change at Cycle 6 Day 1 - Dyspnoea | 0.38 (17.86) | 0.40 (21.64)
  Baseline - Insomnia: number analyzed (Participants) | 97 | 96
  Baseline - Insomnia | 25.09 (27.23) | 28.13 (32.92)
  Change at Cycle 1 Day 1 - Insomnia: number analyzed (Participants) | 89 | 91
  Change at Cycle 1 Day 1 - Insomnia | -1.12 (27.27) | 4.40 (31.51)
  Change at Cycle 3 Day 1 - Insomnia: number analyzed (Participants) | 88 | 89
  Change at Cycle 3 Day 1 - Insomnia | 0.00 (27.68) | -3.00 (34.68)
  Change at Cycle 6 Day 1 - Insomnia: number analyzed (Participants) | 88 | 84
  Change at Cycle 6 Day 1 - Insomnia | 0.76 (28.58) | 0.00 (37.67)
  Baseline - Appetite loss: number analyzed (Participants) | 97 | 96
  Baseline - Appetite loss | 10.65 (18.35) | 11.81 (21.07)
  Change at Cycle 1 Day 1 - Appetite loss: number analyzed (Participants) | 88 | 91
  Change at Cycle 1 Day 1 - Appetite loss | 2.27 (27.59) | 2.56 (29.07)
  Change at Cycle 3 Day 1 - Appetite loss: number analyzed (Participants) | 88 | 89
  Change at Cycle 3 Day 1 - Appetite loss | -0.38 (25.01) | 0.00 (25.62)
  Change at Cycle 6 Day 1 - Appetite loss: number analyzed (Participants) | 88 | 84
  Change at Cycle 6 Day 1 - Appetite loss | -1.14 (24.47) | 0.00 (25.87)
  Baseline - Constipation: number analyzed (Participants) | 97 | 96
  Baseline - Constipation | 13.75 (22.95) | 13.89 (22.51)
  Change at Cycle 1 Day 1 - Constipation: number analyzed (Participants) | 89 | 91
  Change at Cycle 1 Day 1 - Constipation | -2.62 (21.45) | 0.00 (19.25)
  Change at Cycle 3 Day 1 - Constipation: number analyzed (Participants) | 88 | 89
  Change at Cycle 3 Day 1 - Constipation | -4.92 (23.99) | 0.00 (25.62)
  Change at Cycle 6 Day 1 - Constipation: number analyzed (Participants) | 88 | 84
  Change at Cycle 6 Day 1 - Constipation | -3.79 (27.88) | 1.98 (21.55)
  Baseline - Diarrhoea: number analyzed (Participants) | 97 | 96
  Baseline - Diarrhoea | 12.37 (25.15) | 12.15 (22.75)
  Change at Cycle 1 Day 1 - Diarrhoea: number analyzed (Participants) | 88 | 91
  Change at Cycle 1 Day 1 - Diarrhoea | 0.00 (26.74) | 4.76 (33.17)
  Change at Cycle 3 Day 1 - Diarrhoea: number analyzed (Participants) | 88 | 89
  Change at Cycle 3 Day 1 - Diarrhoea | -0.38 (24.50) | 2.25 (32.10)
  Change at Cycle 6 Day 1 - Diarrhoea: number analyzed (Participants) | 88 | 84
  Change at Cycle 6 Day 1 - Diarrhoea | 1.89 (29.62) | 4.76 (32.37)
  Baseline - Financial difficulties: number analyzed (Participants) | 97 | 96
  Baseline - Financial difficulties | 28.18 (34.14) | 32.29 (34.35)
  Change at Cycle 1 Day 1 - Financial Difficulties: number analyzed (Participants) | 89 | 91
  Change at Cycle 1 Day 1 - Financial Difficulties | -6.37 (24.04) | -4.40 (28.20)
  Change at Cycle 3 Day 1 - Financial Difficulties: number analyzed (Participants) | 88 | 89
  Change at Cycle 3 Day 1 - Financial Difficulties | -4.92 (27.00) | -6.37 (29.68)
  Change at Cycle 6 Day 1 - Financial Difficulties: number analyzed (Participants) | 88 | 84
  Change at Cycle 6 Day 1 - Financial Difficulties | -2.65 (27.32) | -6.35 (30.82)

13. Secondary Outcome: Adjuvant Cross-over Period: Percentage of HCPs by Their Responses to Questions 1a and 1c of the HCPQ - Drug Preparation Area
Description: HCP was defined as any personnel involved in the drug preparation and/or drug administration processes. HCPs who have had experience with preparation and/or administration of PH FDC SC completed the following questions of the HCPQ: Q1a: Where was the treatment prepared? Q1c: Which healthcare professionals were involved in the treatment preparation processes? The 4 available response options for Q1a were: Participant's home, Hospital pharmacy, Day oncology unit, or Other. The 5 available response options for Q1c were: Physician, Nurse, Pharmacist, All of them or Other. Percentages were rounded off.
Time Frame: Day 1 of Cycles 3 and 6 (Cycle length = 21 days)
Population: Overall number analyzed is the number of HCPs who answered Q1a and Q1c of the HCPQ. Number analyzed is the number of HCPs who answered Q1a and Q1c of the HCPQ at the specified timepoint.
Measure: Number; unit: percentage of HCPs
Arm/Group | Arm C, Adjuvant Cross-over Phase: PH FDC SC in Hospital, Then at Home | Arm D, Adjuvant Cross-Over Phase: PH FDC SC at Home, Then in Hospital
Number analyzed (Participants) | 78 | 77
percentage of HCPs
  Cycle 3 Day 1: Q1a: Participant's Home: number analyzed (Participants) | 62 | 64
  Cycle 3 Day 1: Q1a: Participant's Home | 0 | 90.6
  Cycle 3 Day 1: Q1a: Hospital Pharmacy: number analyzed (Participants) | 62 | 64
  Cycle 3 Day 1: Q1a: Hospital Pharmacy | 72.6 | 9.4
  Cycle 3 Day 1: Q1a: Day Oncology Unit: number analyzed (Participants) | 62 | 64
  Cycle 3 Day 1: Q1a: Day Oncology Unit | 17.7 | 0
  Cycle 3 Day 1: Q1a: Other: number analyzed (Participants) | 62 | 64
  Cycle 3 Day 1: Q1a: Other | 9.7 | 0
  Cycle 3 Day 1: Q1c: Physician: number analyzed (Participants) | 77 | 77
  Cycle 3 Day 1: Q1c: Physician | 0 | 11.7
  Cycle 3 Day 1: Q1c: Nurse: number analyzed (Participants) | 77 | 77
  Cycle 3 Day 1: Q1c: Nurse | 35.1 | 75.3
  Cycle 3 Day 1: Q1c: Pharmacist: number analyzed (Participants) | 77 | 77
  Cycle 3 Day 1: Q1c: Pharmacist | 59.7 | 7.8
  Cycle 3 Day 1: Q1c: All of Them: number analyzed (Participants) | 77 | 77
  Cycle 3 Day 1: Q1c: All of Them | 2.6 | 2.6
  Cycle 3 Day 1: Q1c: Other: number analyzed (Participants) | 77 | 77
  Cycle 3 Day 1: Q1c: Other | 2.6 | 2.6
  Cycle 6 Day 1: Q1a: Participant's Home: number analyzed (Participants) | 63 | 67
  Cycle 6 Day 1: Q1a: Participant's Home | 95.2 | 0
  Cycle 6 Day 1: Q1a: Hospital Pharmacy: number analyzed (Participants) | 63 | 67
  Cycle 6 Day 1: Q1a: Hospital Pharmacy | 4.8 | 71.6
  Cycle 6: Q1a: Day Oncology Unit: number analyzed (Participants) | 63 | 67
  Cycle 6: Q1a: Day Oncology Unit | 0 | 20.9
  Cycle 6 Day 1: Q1a: Other: number analyzed (Participants) | 63 | 67
  Cycle 6 Day 1: Q1a: Other | 0 | 7.5
  Cycle 6 Day 1: Q1c: Physician: number analyzed (Participants) | 78 | 72
  Cycle 6 Day 1: Q1c: Physician | 5.1 | 2.8
  Cycle 6 Day 1: Q1c: Nurse: number analyzed (Participants) | 78 | 72
  Cycle 6 Day 1: Q1c: Nurse | 88.5 | 29.2
  Cycle 6 Day 1: Q1c: Pharmacist: number analyzed (Participants) | 78 | 72
  Cycle 6 Day 1: Q1c: Pharmacist | 2.6 | 58.3
  Cycle 6 Day 1: Q1c: All of them: number analyzed (Participants) | 78 | 72
  Cycle 6 Day 1: Q1c: All of them | 2.6 | 5.6
  Cycle 6 Day 1: Q1c: Other: number analyzed (Participants) | 78 | 72
  Cycle 6 Day 1: Q1c: Other | 1.3 | 4.2

14. Secondary Outcome: Adjuvant Cross-over Period: Duration of Treatment Preparation, According to HCPs' Responses to Question 1b of the HCPQ - Drug Preparation Area
Description: HCP was defined as any personnel involved in the drug preparation and/or drug administration processes. HCPs who have had experience with preparation and/or administration of PH FDC SC completed the following parts of question Q1b: Q1b(1): How long did it take to prepare the treatment for use? Q1b(2): Time from the preparation place to reach the participant's home.
Time Frame: Day 1 of Cycles 3 and 6 (Cycle length = 21 days)
Population: Overall number analyzed is the number of HCPs who answered Q1b of the HCPQ. Number analyzed is the number of HCPs who answered Q1b of the HCPQ at the specified timepoint.
Measure: Median (Full Range); unit: minutes
Arm/Group | Arm C, Adjuvant Cross-over Phase: PH FDC SC in Hospital, Then at Home | Arm D, Adjuvant Cross-Over Phase: PH FDC SC at Home, Then in Hospital
Number analyzed (Participants) | 20 | 19
minutes
  Cycle 3 Day 1: Q1b(1) | 5.0 [1 to 33] | 5.0 [1 to 30]
  Cycle 3 Day 1: Q1b(2): number analyzed (Participants) | 7 | 16
  Cycle 3 Day 1: Q1b(2) | 5.0 [0 to 35] | 1.0 [0 to 70]
  Cycle 6 Day 1: Q1b(1): number analyzed (Participants) | 18 | 9
  Cycle 6 Day 1: Q1b(1) | 5.0 [1 to 30] | 4.0 [1 to 15]
  Cycle 6 Day 1: Q1b(2): number analyzed (Participants) | 15 | 7
  Cycle 6 Day 1: Q1b(2) | 0.0 [0 to 60] | 3.0 [0 to 30]

15. Secondary Outcome: Adjuvant Cross-over Period: Percentage of HCPs by Their Responses to Questions 2, 3 and 4 of the HCPQ - Drug Preparation Area
Description: HCP was defined as any personnel involved in the drug preparation and/or drug administration processes. HCPs who have had experience with preparation and/or administration of PH FDC SC completed the questions 2, 3 and 4 of the HCPQ: Q2: If all PH FDC SC injections were switched from an in-hospital setting to the participant´s home, please indicate how strongly you agree or disagree with each of the following statements: 2a: Staff will have increased availability for other tasks in the hospital´s pharmacy. 2b: Administrative procedures related to PH FDC SC will require less time. 2c: Number of preparation steps and staff time commitment are reduced. The 5 response options were: Strongly disagree, Disagree, Neutral, Agree, Strongly agree or Not applicable. Q3: Which took less time? Q4: Which required less use of institutional resources? The 4 available options were: Participant's home, In hospital, No difference, or Unsure. Percentages were rounded off.
Time Frame: Day 1 of Cycle 6 (Cycle length = 21 days)
Population: Overall number analyzed is the number of HCPs who answered any of the questions Q2, Q3, and Q4 of the HCPQ. Number analyzed is the number of HCPs who answered each sub-question of Q2, and Q3, and Q4 of the HCPQ.
Measure: Number; unit: percentage of HCPs
Arm/Group | Arm C, Adjuvant Cross-over Phase: PH FDC SC in Hospital, Then at Home | Arm D, Adjuvant Cross-Over Phase: PH FDC SC at Home, Then in Hospital
Number analyzed (Participants) | 81 | 75
percentage of HCPs
  Q2a: Strongly Disagree | 2.5 | 1.3
  Q2a: Disagree | 0 | 18.7
  Q2a: Neutral | 6.2 | 16.0
  Q2a: Agree | 43.2 | 21.3
  Q2a: Strongly Agree | 38.3 | 37.3
  Q2a: Not Applicable | 9.9 | 5.3
  Q2b: Strongly Disagree: number analyzed (Participants) | 81 | 74
  Q2b: Strongly Disagree | 4.9 | 2.7
  Q2b: Disagree: number analyzed (Participants) | 81 | 74
  Q2b: Disagree | 2.5 | 24.3
  Q2b: Neutral: number analyzed (Participants) | 81 | 74
  Q2b: Neutral | 13.6 | 13.5
  Q2b: Agree: number analyzed (Participants) | 81 | 74
  Q2b: Agree | 33.3 | 18.9
  Q2b: Strongly Agree: number analyzed (Participants) | 81 | 74
  Q2b: Strongly Agree | 35.8 | 35.1
  Q2b: Not Applicable: number analyzed (Participants) | 81 | 74
  Q2b: Not Applicable | 9.9 | 5.4
  Q2c: Strongly Disagree: number analyzed (Participants) | 81 | 74
  Q2c: Strongly Disagree | 2.5 | 0
  Q2c: Disagree: number analyzed (Participants) | 81 | 74
  Q2c: Disagree | 2.5 | 18.9
  Q2c: Neutral: number analyzed (Participants) | 81 | 74
  Q2c: Neutral | 6.2 | 21.6
  Q2c: Agree: number analyzed (Participants) | 81 | 74
  Q2c: Agree | 39.5 | 16.2
  Q2c: Strongly Agree: number analyzed (Participants) | 81 | 74
  Q2c: Strongly Agree | 38.3 | 37.8
  Q2c: Not Applicable: number analyzed (Participants) | 81 | 74
  Q2c: Not Applicable | 11.1 | 5.4
  Q3: Participant's Home: number analyzed (Participants) | 79 | 72
  Q3: Participant's Home | 59.5 | 22.2
  Q3: In hospital: number analyzed (Participants) | 79 | 72
  Q3: In hospital | 2.5 | 36.1
  Q3: No Difference: number analyzed (Participants) | 79 | 72
  Q3: No Difference | 11.4 | 31.9
  Q3: Unsure: number analyzed (Participants) | 79 | 72
  Q3: Unsure | 26.6 | 9.7
  Q4: Participant's Home: number analyzed (Participants) | 79 | 72
  Q4: Participant's Home | 73.4 | 38.9
  Q4: In hospital: number analyzed (Participants) | 79 | 72
  Q4: In hospital | 5.1 | 36.1
  Q4: No Difference: number analyzed (Participants) | 79 | 72
  Q4: No Difference | 8.9 | 19.4
  Q4: Unsure: number analyzed (Participants) | 79 | 72
  Q4: Unsure | 12.7 | 5.6

16. Secondary Outcome: Adjuvant Cross-over Period: Duration of Administering Treatment, According to HCPs' Responses to Question 1a to 1f of the HCPQ - Administering Treatment
Description: HCP was defined as any personnel involved in the drug preparation and/or drug administration processes. HCPs who have had experience with the preparation and/or administration of PH FDC SC completed the following questions of the HCPQ: Q1a: How long did it take to travel to the participant's home to administer PH FDC SC? Q1b: How long did it take for the participant to travel to the hospital to receive PH FDC SC? Q1c: How long did it take to administer PH FDC SC? Q1d: How long was the participant treatment time? Q1e: How much time did the participant spend in hospital? Q1f: How much time did you spend at the participant's home? From arrival to departure time.
Time Frame: Day 1 of Cycles 3 and 6 (Cycle length = 21 days)
Population: Overall number analyzed is the number of HCPs who answered Q1a to Q1f of the HCPQ. Number analyzed is the number of HCPs who answered Q1a to Q1f of the HCPQ at the specified timepoint.
Measure: Median (Full Range); unit: minutes
Arm/Group | Arm C, Adjuvant Cross-over Phase: PH FDC SC in Hospital, Then at Home | Arm D, Adjuvant Cross-Over Phase: PH FDC SC at Home, Then in Hospital
Number analyzed (Participants) | 81 | 76
minutes
  Cycle 3 Day 1: Q1a: number analyzed (Participants) | 2 | 73
  Cycle 3 Day 1: Q1a | 82.5 [60 to 105] | 60.0 [11 to 540]
  Cycle 3 Day 1: Q1b: number analyzed (Participants) | 67 | 23
  Cycle 3 Day 1: Q1b | 60.0 [10 to 420] | 60.0 [10 to 660]
  Cycle 3 Day 1: Q1c: number analyzed (Participants) | 75 | 76
  Cycle 3 Day 1: Q1c | 5.0 [5 to 13] | 5.0 [5 to 30]
  Cycle 3 Day 1: Q1d: number analyzed (Participants) | 75 | 75
  Cycle 3 Day 1: Q1d | 30.0 [5 to 540] | 75.0 [5 to 240]
  Cycle 3 Day 1: Q1e: number analyzed (Participants) | 73 | 14
  Cycle 3 Day 1: Q1e | 120.0 [25 to 586] | 180.0 [70 to 360]
  Cycle 3 Day 1: Q1f: number analyzed (Participants) | 0 | 69
  Cycle 3 Day 1: Q1f |  | 90.0 [40 to 175]
  Cycle 6 Day 1: Q1a: number analyzed (Participants) | 80 | 4
  Cycle 6 Day 1: Q1a | 65.0 [5 to 480] | 85.0 [50 to 180]
  Cycle 6 Day 1: Q1b: number analyzed (Participants) | 35 | 71
  Cycle 6 Day 1: Q1b | 60.0 [15 to 480] | 60.0 [5 to 660]
  Cycle 6 Day 1: Q1c: number analyzed (Participants) | 81 | 74
  Cycle 6 Day 1: Q1c | 5.0 [5 to 30] | 5.0 [5 to 10]
  Cycle 6 Day 1: Q1d: number analyzed (Participants) | 81 | 73
  Cycle 6 Day 1: Q1d | 90.0 [8 to 165] | 30.0 [5 to 240]
  Cycle 6 Day 1: Q1e: number analyzed (Participants) | 27 | 74
  Cycle 6 Day 1: Q1e | 120.0 [50 to 600] | 120.0 [25 to 480]
  Cycle 6 Day 1: Q1f: number analyzed (Participants) | 79 | 1
  Cycle 6 Day 1: Q1f | 90.0 [20 to 165] | 90.0 [90 to 90]

17. Secondary Outcome: Adjuvant Cross-over Period: Percentage of HCPs by Their Responses to Questions 1g, 1h, and 1i of the HCPQ - Administering Treatment
Description: HCP was defined as any personnel involved in the drug preparation and/or drug administration processes. HCPs who have had experience with the preparation and/or administration of PH FDC SC completed the following questions of the HCPQ: Q1g. Does the participant still have implanted IV access? The 2 available responses were: Yes or No. Q1h: If question 1g was answered 'No', when was the IV access removed? The 3 available responses were: After surgery and before initiating adjuvant treatment; After initiating adjuvant treatment, or Not applicable. Q1i: If question 1g was answered 'Yes', what is the main reason to keep the IV access? The 5 available responses were: Local protocol; Risk of recurrence; Participant preference; Not applicable, or Other. Percentages were rounded off.
Time Frame: Day 1 of Cycles 3 and 6 (Cycle length = 21 days)
Population: Overall number analyzed is the number of HCPs who answered Q1g to Q1i of the HCPQ. Number analyzed is the number of HCPs who answered Q1g to Q1i of the HCPQ at the specified timepoint.
Measure: Number; unit: percentage of HCPs
Arm/Group | Arm C, Adjuvant Cross-over Phase: PH FDC SC in Hospital, Then at Home | Arm D, Adjuvant Cross-Over Phase: PH FDC SC at Home, Then in Hospital
Number analyzed (Participants) | 59 | 61
percentage of HCPs
  Cycle 3 Day 1: Q1g: Yes: number analyzed (Participants) | 45 | 55
  Cycle 3 Day 1: Q1g: Yes | 35.6 | 14.5
  Cycle 3 Day 1: Q1g: No: number analyzed (Participants) | 45 | 55
  Cycle 3 Day 1: Q1g: No | 64.4 | 85.5
  Cycle 3 Day 1: Q1h: After Surgery and Before Adjuvant Treatment: number analyzed (Participants) | 28 | 47
  Cycle 3 Day 1: Q1h: After Surgery and Before Adjuvant Treatment | 7.1 | 4.3
  Cycle 3 Day 1: Q1h: After Initiating Adjuvant Treatment: number analyzed (Participants) | 28 | 47
  Cycle 3 Day 1: Q1h: After Initiating Adjuvant Treatment | 7.1 | 10.6
  Cycle 3 Day 1: Q1h: Not Applicable: number analyzed (Participants) | 28 | 47
  Cycle 3 Day 1: Q1h: Not Applicable | 85.7 | 85.1
  Cycle 3 Day 1: Q1i: Local Protocol: number analyzed (Participants) | 20 | 14
  Cycle 3 Day 1: Q1i: Local Protocol | 45.0 | 21.4
  Cycle 3 Day 1: Q1i: Risk of Recurrence: number analyzed (Participants) | 20 | 14
  Cycle 3 Day 1: Q1i: Risk of Recurrence | 10.0 | 14.3
  Cycle 3 Day 1: Q1i: Participant Preference: number analyzed (Participants) | 20 | 14
  Cycle 3 Day 1: Q1i: Participant Preference | 25.0 | 14.3
  Cycle 3 Day 1: Q1i: Not Applicable: number analyzed (Participants) | 20 | 14
  Cycle 3 Day 1: Q1i: Not Applicable | 15.0 | 50.0
  Cycle 3 Day 1: Q1i: Other: number analyzed (Participants) | 20 | 14
  Cycle 3 Day 1: Q1i: Other | 5.0 | 0
  Cycle 6 Day 1: Q1g: Yes | 23.7 | 23.0
  Cycle 6 Day 1: Q1g: No | 76.3 | 77.0
  Cycle 6 Day 1: Q1h: After Surgery and Before Adjuvant Treatment: number analyzed (Participants) | 48 | 47
  Cycle 6 Day 1: Q1h: After Surgery and Before Adjuvant Treatment | 10.4 | 6.4
  Cycle 6 Day 1: Q1h: After Initiating Adjuvant Treatment: number analyzed (Participants) | 48 | 47
  Cycle 6 Day 1: Q1h: After Initiating Adjuvant Treatment | 0 | 6.4
  Cycle 6 Day 1: Q1h: Not Applicable: number analyzed (Participants) | 48 | 47
  Cycle 6 Day 1: Q1h: Not Applicable | 89.6 | 87.2
  Cycle 6 Day 1: Q1i: Local Protocol: number analyzed (Participants) | 29 | 21
  Cycle 6 Day 1: Q1i: Local Protocol | 27.6 | 42.9
  Cycle 6 Day 1: Q1i: Risk of Recurrence: number analyzed (Participants) | 29 | 21
  Cycle 6 Day 1: Q1i: Risk of Recurrence | 3.4 | 4.8
  Cycle 6 Day 1: Q1i: Participant Preference: number analyzed (Participants) | 29 | 21
  Cycle 6 Day 1: Q1i: Participant Preference | 13.8 | 4.8
  Cycle 6 Day 1: Q1i: Not Applicable: number analyzed (Participants) | 29 | 21
  Cycle 6 Day 1: Q1i: Not Applicable | 51.7 | 38.1
  Cycle 6 Day 1: Q1i: Other: number analyzed (Participants) | 29 | 21
  Cycle 6 Day 1: Q1i: Other | 3.4 | 9.5

18. Secondary Outcome: Adjuvant Cross-over Period: Percentage of HCPs by Their Responses to Questions 1j, 1k, and 1l of the HCPQ - Administering Treatment
Description: HCPs who have had experience with the preparation and/or administration of PH FDC SC completed the following questions of the HCPQ: Q1j: How long do you keep implanted IV access in early human epidermal growth factor receptor 2 (HER2)-positive breast cancer participants with pCR following surgery in your institution? The 5 available responses were: <12 months, ≥12 months, 18 months, <24 months, ≥24 months. Q1k: When is the decision point for you to decide to remove IV access for early HER2+ breast cancer participants? The 6 available responses were: Before surgery, After surgery, After PCR results, After completion of full adjuvant therapy, After completion of IV antineoplastic within adjuvant therapy, and Other. Q1l: Do you consider it necessary to keep implanted IV access knowing that the participant's treatment will be SC until the full 18 cycles? The 3 available responses were: Yes, No, and Unsure. Percentages were rounded off.
Time Frame: Day 1 of Cycle 6 (Cycle length = 21 days)
Population: Overall number analyzed is the number of HCPs who answered any of the questions from Q1j to Q1l of the HCPQ. Number analyzed is the number of HCPs who answered each specific question (Q1j to Q1l) of the HCPQ.
Measure: Number; unit: percentage of HCPs
Arm/Group | Arm C, Adjuvant Cross-over Phase: PH FDC SC in Hospital, Then at Home | Arm D, Adjuvant Cross-Over Phase: PH FDC SC at Home, Then in Hospital
Number analyzed (Participants) | 44 | 43
percentage of HCPs
  Q1j: <12 Months: number analyzed (Participants) | 28 | 37
  Q1j: <12 Months | 10.7 | 27.0
  Q1j: ≥12 Months: number analyzed (Participants) | 28 | 37
  Q1j: ≥12 Months | 28.6 | 16.2
  Q1j: 18 Months: number analyzed (Participants) | 28 | 37
  Q1j: 18 Months | 14.3 | 16.2
  Q1j: <24 Months: number analyzed (Participants) | 28 | 37
  Q1j: <24 Months | 3.6 | 8.1
  Q1j: ≥24 Months: number analyzed (Participants) | 28 | 37
  Q1j: ≥24 Months | 42.9 | 32.4
  Q1k: Before Surgery: number analyzed (Participants) | 44 | 39
  Q1k: Before Surgery | 0 | 2.6
  Q1k: After Surgery: number analyzed (Participants) | 44 | 39
  Q1k: After Surgery | 2.3 | 10.3
  Q1k: After PCR Results: number analyzed (Participants) | 44 | 39
  Q1k: After PCR Results | 15.9 | 20.5
  Q1k: After Completion of Full Adjuvant Therapy: number analyzed (Participants) | 44 | 39
  Q1k: After Completion of Full Adjuvant Therapy | 15.9 | 28.2
  Q1k: After Completion of IV Antineoplastic Within Adjuvant Therapy: number analyzed (Participants) | 44 | 39
  Q1k: After Completion of IV Antineoplastic Within Adjuvant Therapy | 29.5 | 5.1
  Q1k: Other: number analyzed (Participants) | 44 | 39
  Q1k: Other | 36.4 | 33.3
  Q1l: Yes: number analyzed (Participants) | 42 | 43
  Q1l: Yes | 11.9 | 37.2
  Q1l: No: number analyzed (Participants) | 42 | 43
  Q1l: No | 35.7 | 37.2
  Q1l: Unsure: number analyzed (Participants) | 42 | 43
  Q1l: Unsure | 52.4 | 25.6

19. Secondary Outcome: Adjuvant Cross-over Period: Percentage of HCPs by Their Responses to Question 2 of the HCPQ - Administering Treatment
Description: HCPs who have had experience with the preparation and/or administration of PH FDC SC completed the following question of the HCPQ: Q2: If all PH FDC SC injections were switched from an in-hospital setting to the participant's home, please indicate how strongly you agree/disagree with each of the following statements: 2a: PH FDC SC's SC route of administration allows for more flexible treatment scheduling. 2b: Frees up infusion chairs or outpatient procedure rooms used to administer SC injections. 2c: Waiting list for infusion chairs or outpatient procedure rooms is reduced. 2d: Staff's work burden is reduced, enhancing work performance. 2e: More interaction time between HCPs and participants on IV treatment. 2f: Staff has more time for administrative tasks. 2g: Participants will spend less time in hospital. 2h: Participants prefer PH FDC SC at home. The 6 available responses were: Strongly disagree, Disagree, Neutral, Agree, Strongly agree, & Not applicable.
Time Frame: Day 1 of Cycle 6 (Cycle length = 21 days)
Population: Overall number analyzed is the number of HCPs who answered Q2 of the HCPQ. Number analyzed is the number of HCPs who answered each sub-question of Q2 (Q2a-Q2h) of the HCPQ. Percentages were rounded off.
Measure: Number; unit: percentage of HCPs
Arm/Group | Arm C, Adjuvant Cross-over Phase: PH FDC SC in Hospital, Then at Home | Arm D, Adjuvant Cross-Over Phase: PH FDC SC at Home, Then in Hospital
Number analyzed (Participants) | 79 | 75
percentage of HCPs
  Q2a: Strongly Disagree | 6.3 | 0
  Q2a: Disagree | 0 | 1.3
  Q2a: Neutral | 6.3 | 8.0
  Q2a: Agree | 30.4 | 41.3
  Q2a: Strongly Agree | 55.7 | 45.3
  Q2a: Not Applicable | 1.3 | 4.0
  Q2b: Strongly Disagree: number analyzed (Participants) | 78 | 75
  Q2b: Strongly Disagree | 6.4 | 1.3
  Q2b: Disagree: number analyzed (Participants) | 78 | 75
  Q2b: Disagree | 0 | 5.3
  Q2b: Neutral: number analyzed (Participants) | 78 | 75
  Q2b: Neutral | 7.7 | 6.7
  Q2b: Agree: number analyzed (Participants) | 78 | 75
  Q2b: Agree | 29.5 | 33.3
  Q2b: Strongly Agree: number analyzed (Participants) | 78 | 75
  Q2b: Strongly Agree | 55.1 | 49.3
  Q2b: Not Applicable: number analyzed (Participants) | 78 | 75
  Q2b: Not Applicable | 1.3 | 4.0
  Q2c: Strongly Disagree: number analyzed (Participants) | 78 | 75
  Q2c: Strongly Disagree | 7.7 | 2.7
  Q2c: Disagree: number analyzed (Participants) | 78 | 75
  Q2c: Disagree | 0 | 1.3
  Q2c: Neutral: number analyzed (Participants) | 78 | 75
  Q2c: Neutral | 0 | 5.3
  Q2c: Agree: number analyzed (Participants) | 78 | 75
  Q2c: Agree | 33.3 | 33.3
  Q2c: Strongly Agree: number analyzed (Participants) | 78 | 75
  Q2c: Strongly Agree | 57.7 | 53.3
  Q2c: Not Applicable: number analyzed (Participants) | 78 | 75
  Q2c: Not Applicable | 1.3 | 4.0
  Q2d: Strongly Disagree: number analyzed (Participants) | 77 | 75
  Q2d: Strongly Disagree | 6.5 | 0
  Q2d: Disagree: number analyzed (Participants) | 77 | 75
  Q2d: Disagree | 3.9 | 9.3
  Q2d: Neutral: number analyzed (Participants) | 77 | 75
  Q2d: Neutral | 14.3 | 14.7
  Q2d: Agree: number analyzed (Participants) | 77 | 75
  Q2d: Agree | 27.3 | 25.3
  Q2d: Strongly Agree: number analyzed (Participants) | 77 | 75
  Q2d: Strongly Agree | 46.8 | 42.7
  Q2d: Not Applicable: number analyzed (Participants) | 77 | 75
  Q2d: Not Applicable | 1.3 | 8.0
  Q2e: Strongly Disagree: number analyzed (Participants) | 78 | 75
  Q2e: Strongly Disagree | 6.4 | 0
  Q2e: Disagree: number analyzed (Participants) | 78 | 75
  Q2e: Disagree | 2.6 | 2.7
  Q2e: Neutral: number analyzed (Participants) | 78 | 75
  Q2e: Neutral | 19.2 | 20.0
  Q2e: Agree: number analyzed (Participants) | 78 | 75
  Q2e: Agree | 26.9 | 33.3
  Q2e: Strongly Agree: number analyzed (Participants) | 78 | 75
  Q2e: Strongly Agree | 43.6 | 33.3
  Q2e: Not Applicable: number analyzed (Participants) | 78 | 75
  Q2e: Not Applicable | 1.3 | 10.7
  Q2f: Strongly Disagree: number analyzed (Participants) | 78 | 75
  Q2f: Strongly Disagree | 7.7 | 0
  Q2f: Disagree: number analyzed (Participants) | 78 | 75
  Q2f: Disagree | 2.6 | 4.0
  Q2f: Neutral: number analyzed (Participants) | 78 | 75
  Q2f: Neutral | 9.0 | 25.3
  Q2f: Agree: number analyzed (Participants) | 78 | 75
  Q2f: Agree | 32.1 | 22.7
  Q2f: Strongly Agree: number analyzed (Participants) | 78 | 75
  Q2f: Strongly Agree | 47.4 | 40.0
  Q2f: Not Applicable: number analyzed (Participants) | 78 | 75
  Q2f: Not Applicable | 1.3 | 8.0
  Q2g: Strongly Disagree: number analyzed (Participants) | 78 | 75
  Q2g: Strongly Disagree | 6.4 | 0
  Q2g: Disagree: number analyzed (Participants) | 78 | 75
  Q2g: Disagree | 0 | 1.3
  Q2g: Neutral: number analyzed (Participants) | 78 | 75
  Q2g: Neutral | 0 | 6.7
  Q2g: Agree: number analyzed (Participants) | 78 | 75
  Q2g: Agree | 24.4 | 32.0
  Q2g: Strongly Agree: number analyzed (Participants) | 78 | 75
  Q2g: Strongly Agree | 67.9 | 56.0
  Q2g: Not Applicable: number analyzed (Participants) | 78 | 75
  Q2g: Not Applicable | 1.3 | 4.0
  Q2h: Strongly Disagree: number analyzed (Participants) | 77 | 75
  Q2h: Strongly Disagree | 6.5 | 2.7
  Q2h: Disagree: number analyzed (Participants) | 77 | 75
  Q2h: Disagree | 3.9 | 18.7
  Q2h: Neutral: number analyzed (Participants) | 77 | 75
  Q2h: Neutral | 15.6 | 28.0
  Q2h: Agree: number analyzed (Participants) | 77 | 75
  Q2h: Agree | 23.4 | 17.3
  Q2h: Strongly Agree: number analyzed (Participants) | 77 | 75
  Q2h: Strongly Agree | 49.4 | 29.3
  Q2h: Not Applicable: number analyzed (Participants) | 77 | 75
  Q2h: Not Applicable | 1.3 | 4.0

20. Secondary Outcome: Adjuvant Cross-over Period: Percentage of HCPs by Their Responses to Questions 3 to 7 of the HCPQ - Administering Treatment
Description: HCP was defined as any personnel involved in the drug preparation and/or drug administration processes. HCPs who have had experience with the preparation and/or administration of PH FDC SC completed the following questions of the HCPQ: Q3: Which was more convenient for the participant? Q4: Which was better for optimising participant care? Q5: Which required less use of institutional resources? Q6: Which was preferred by participants? The 4 responses available were: Participant's home, In hospital, No difference, and Unsure. Q7: How frequently would you recommend PH FDC SC at home to your participants in the future? The 3 responses available were: Always, Sometimes, and Never. Percentages were rounded off.
Time Frame: Day 1 of Cycle 6 (Cycle length = 21 days)
Population: Overall number analyzed is the number of HCPs who answered any of the questions from Q3 to Q7 of the HCPQ. Number analyzed is the number of HCPs who answered each specific question (Q3 to Q7) of the HCPQ.
Measure: Number; unit: percentage of HCPs
Arm/Group | Arm C, Adjuvant Cross-over Phase: PH FDC SC in Hospital, Then at Home | Arm D, Adjuvant Cross-Over Phase: PH FDC SC at Home, Then in Hospital
Number analyzed (Participants) | 81 | 74
percentage of HCPs
  Q3: Participant's Home | 84.0 | 45.9
  Q3: In Hospital | 7.4 | 40.5
  Q3: No Difference | 6.2 | 6.8
  Q3: Unsure | 2.5 | 6.8
  Q4: Participant's Home | 80.2 | 28.4
  Q4: In Hospital | 7.4 | 52.7
  Q4: No Difference | 6.2 | 12.2
  Q4: Unsure | 6.2 | 6.8
  Q5: Participant's Home | 67.9 | 40.5
  Q5: In Hospital | 6.2 | 27.0
  Q5: No Difference | 17.3 | 16.2
  Q5: Unsure | 8.6 | 16.2
  Q6: Participant's Home | 79.0 | 41.9
  Q6: In Hospital | 11.1 | 44.6
  Q6: No Difference | 6.2 | 6.8
  Q6: Unsure | 3.7 | 6.8
  Q7: Always: number analyzed (Participants) | 81 | 73
  Q7: Always | 80.2 | 43.8
  Q7: Sometimes: number analyzed (Participants) | 81 | 73
  Q7: Sometimes | 17.3 | 43.8
  Q7: Never: number analyzed (Participants) | 81 | 73
  Q7: Never | 2.5 | 12.3

21. Secondary Outcome: Adjuvant Phase: HRQoL Assessed by EORTC QLQ C30 Scores in Participants Treated With Trastuzumab Emtansine IV
Description: as for outcome 12
Time Frame: Day 1 of Cycles 1 and 6 (1 Cycle = 21 days)
Reporting Status: Not Posted

22. Secondary Outcome: Percentage of Participants Who Selected the Administration of PH FDC SC in the Home Setting Compared With the Hospital Setting in the Treatment Continuation Period
Description: The percentage of participants who chose to receive PH FDC SC in the home setting or in the hospital setting during the treatment continuation period is reported.
Time Frame: Upon completion of adjuvant cross-over period (Day 1 of Cycle 8 or 9; Cycle length = 21 days)
Population: The analysis includes all randomized participants assigned into the cross-over period who received at least one dose of PH FDC SC and entered the treatment continuation phase.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm C, Adjuvant Cross-over Phase: PH FDC SC in Hospital, Then at Home | Arm D, Adjuvant Cross-Over Phase: PH FDC SC at Home, Then in Hospital
Number analyzed (Participants) | 96 | 92
Percentage of participants
  Choice of Home Setting | 68.8 | 54.3
  Choice of Hospital Setting | 31.2 | 45.7

23. Secondary Outcome: Neoadjuvant Phase: Number of Participants With Adverse Events (AEs), Grade ≥ 3 AEs, Serious AEs (SAEs), and Cardiac AEs
Description: AE was defined as any untoward medical occurrence in a clinical study participant temporally associated with use of a study treatment, whether or not considered related to the study treatment. SAE=any untoward medical occurrence that, at any dose: Results in death; Is life threatening; Requires inpatient hospitalization/prolongation of existing hospitalization; Results in persistent disability/incapacity &/or is a congenital anomaly/birth defect. Cardiac AEs=asymptomatic decline in left ventricular ejection fraction (LVEF) of ≥10% from baseline to an LVEF <50%; asymptomatic decline in LVEF requiring treatment/leading to discontinuation of study treatment; congestive heart failure (CHF). AEs ≥Grade 3=marked limitation of physical activity. Comfortable at rest, but any ordinary activity causes fatigue, palpitation/dyspnea; Inability to carry any physical activity without discomfort. Symptoms of cardiac insufficiency at rest. Any physical activity leads to discomfort.
Time Frame: From initiation of study treatment until 28 days after the last treatment cycle (up to approximately 7.4 months)
Population: Neoadjuvant safety analysis set (SASab) included all randomized participants who received at least one study treatment during the neoadjuvant phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A, Neoadjuvant Phase: P+H IV | Arm B, Neoadjuvant Phase: PH FDC SC
Number analyzed (Participants) | 115 | 228
Participants
  AEs | 113 | 227
  SAEs | 19 | 43
  Grade ≥ 3 AEs | 46 | 103
  Cardiac AEs | 1 | 3

24. Secondary Outcome: Neoadjuvant Phase: Number of Participants With Premature Withdrawal From PH FDC SC and P+H IV Due to AEs
Description: An AE was any untoward medical occurrence in a clinical study participant temporally associated with the use of a study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable & unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study intervention. Participants who discontinued the study due to AEs are reported here.
Time Frame: Up to Cycle 8 (1 Cycle = 21 days)
Population: SASab included all randomized participants who received at least one study treatment during the neoadjuvant phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A, Neoadjuvant Phase: P+H IV | Arm B, Neoadjuvant Phase: PH FDC SC
Number analyzed (Participants) | 115 | 228
Participants | 1 | 8

25. Secondary Outcome: Adjuvant Cross-over Period: Number of Participants With AEs, Grade ≥ 3 AEs, SAEs, and Cardiac AEs
Description: AE was defined as any untoward medical occurrence in a clinical study participant temporally associated with use of a study treatment, whether or not considered related to the study treatment. SAE=any untoward medical occurrence that, at any dose: Results in death; Is life threatening; Requires inpatient hospitalization/prolongation of existing hospitalization; Results in persistent disability/incapacity &/or is a congenital anomaly/birth defect. Cardiac AEs=asymptomatic decline in LVEF of ≥10% from baseline to an LVEF <50%; asymptomatic decline in LVEF requiring treatment/leading to discontinuation of study treatment; CHF. AEs ≥Grade 3=marked limitation of physical activity. Comfortable at rest, but any ordinary activity causes fatigue, palpitation/dyspnea; Inability to carry any physical activity without discomfort. Symptoms of cardiac insufficiency at rest. Any physical activity leads to discomfort.
Time Frame: From initiation of study treatment until 28 days after the last treatment cycle (up to approximately 5.8 months)
Population: Adjuvant safety analysis set (SAScd+) included all participants with pCR who received at least one dose of PH FDC SC during the adjuvant phase. AEs for the cross-over period are pooled per treatment administration setting.
Measure: Count of Participants; unit: Participants
Groups:
- Adjuvant Cross-Over Period: PH FDC SC in Hospital: Participants who completed the run-in period received maintenance doses of pertuzumab, 600 mg, trastuzumab, 600 mg, and rHuPH20, 20,000 U, as a SC injection for 3 cycles in the hospital setting during the cross-over period (Cycle length = 21 days).
- Adjuvant Cross-Over Period: PH FDC SC at Home: Participants who completed the run-in period received maintenance doses of pertuzumab, 600 mg, trastuzumab, 600 mg, and rHuPH20, 20,000 U, as a SC injection for 3 cycles in the home setting during the cross-over period (Cycle length = 21 days).
Arm/Group | Adjuvant Cross-Over Period: PH FDC SC in Hospital | Adjuvant Cross-Over Period: PH FDC SC at Home
Number analyzed (Participants) | 190 | 191
Participants
  AEs | 99 | 89
  SAEs | 1 | 1
  Cardiac AEs | 1 | 2
  Grade ≥3 AEs | 6 | 3

26. Secondary Outcome: Adjuvant Cross-over Period: Number of Participants With Premature Withdrawal From PH FDC SC Due to AEs
Description: as for outcome 24
Time Frame: Up to Cycle 6 (Cycle length = 21 days)
Population: SAScd+ included all participants with pCR who received at least one dose of PH FDC SC during the adjuvant phase. AEs for the cross-over period are pooled per treatment administration setting.
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Cross-Over Period: PH FDC SC in Hospital | Adjuvant Cross-Over Period: PH FDC SC at Home
Number analyzed (Participants) | 190 | 191
Participants | 2 | 2

27. Secondary Outcome: Treatment Continuation Period and Trastuzumab Emtansine IV Period: Number of Participants With AEs, Grade ≥ 3 AEs, SAEs, and Cardiac AEs
Description: as for outcome 25
Time Frame: From initiation of study treatment until 28 days after the last treatment cycle (up to approximately 3.5 years)
Reporting Status: Not Posted

28. Secondary Outcome: Treatment Continuation Period and Trastuzumab Emtansine IV Period: Number of Participants With Premature Withdrawal From PH FDC SC and Trastuzumab Emtansine IV Due to AEs
Description: An AE was any untoward medical occurrence in a clinical study participant temporally associated with the use of a study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable & unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study intervention. Participants who discontinue study due to AEs will be reported.
Time Frame: From initiation of study treatment in the adjuvant phase until 28 days after the last treatment cycle (up to approximately 3.5 years)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From initiation of study treatment until 28 days after the last treatment cycle (Neoadjuvant phase: up to 7.4 months; Adjuvant phase: up to 12.3 months)
Description: SASab=all randomized participants who received at least 1 study treatment during NP. SAScd+=all participants with pCR who received ≥1 dose of PH FDC SC in AP. AEs for cross-over period are pooled per treatment administration setting; some participants discontinued after receiving treatment in 1 setting but not the other. Participants that switched between administration settings during continuation period are counted in both settings. Final AE data will be reported 1 year after study completion.
Groups:
- Adjuvant Cross-Over Phase: PH FDC SC in Hospital: Participants who completed the run-in period received maintenance doses of pertuzumab, 600 mg, trastuzumab, 600 mg, and rHuPH20, 20,000 U, as a SC injection for 3 cycles in the hospital setting during the cross-over period (Cycle length = 21 days).
- Adjuvant Cross-Over Phase: PH FDC SC at Home: Participants who completed the run-in period received maintenance doses of pertuzumab, 600 mg, trastuzumab, 600 mg, and rHuPH20, 20,000 U, as a SC injection for 3 cycles in the home setting during the cross-over period (Cycle length = 21 days).
- Adjuvant Continuation Phase: PH FDC SC in Hospital: Participants who completed the cross-over period and opted to receive further treatment in the hospital setting received maintenance doses of pertuzumab, 600 mg, trastuzumab, 600 mg, and rHuPH20, 20,000 U, as a SC injection up to a maximum of 18 cycles (Cycle length = 21 days).
- Adjuvant Continuation Phase: PH FDC SC at Home: Participants who completed the cross-over period and opted to receive further treatment at home received maintenance doses of pertuzumab, 600 mg, trastuzumab, 600 mg, and rHuPH20, 20,000 U, as a SC injection up to a maximum of 18 cycles (Cycle length = 21 days).
Arm/Group | Arm A, Neoadjuvant Phase: P+H IV | Arm B, Neoadjuvant Phase: PH FDC SC | Adjuvant Run-in Phase: PH FDC SC in Hospital | Adjuvant Cross-Over Phase: PH FDC SC in Hospital | Adjuvant Cross-Over Phase: PH FDC SC at Home | Adjuvant Continuation Phase: PH FDC SC in Hospital | Adjuvant Continuation Phase: PH FDC SC at Home | Arm E, Adjuvant Phase: Trastuzumab Emtansine IV
All-Cause Mortality (participants affected / at risk) | 0/115 | 4/228 | 0/194 | 0/190 | 0/191 | 0/84 | 0/114 | 1/117
Serious Adverse Events (participants affected / at risk) | 19/115 | 43/228 | 3/194 | 1/190 | 1/191 | 1/84 | 0/114 | 9/117
Other Adverse Events (participants affected / at risk) | 113/115 | 222/228 | 84/194 | 77/190 | 64/191 | 26/84 | 31/114 | 107/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A, Neoadjuvant Phase: P+H IV (N=115) | Arm B, Neoadjuvant Phase: PH FDC SC (N=228) | Adjuvant Run-in Phase: PH FDC SC in Hospital (N=194) | Adjuvant Cross-Over Phase: PH FDC SC in Hospital (N=190) | Adjuvant Cross-Over Phase: PH FDC SC at Home (N=191) | Adjuvant Continuation Phase: PH FDC SC in Hospital (N=84) | Adjuvant Continuation Phase: PH FDC SC at Home (N=114) | Arm E, Adjuvant Phase: Trastuzumab Emtansine IV (N=117)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atypical haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 7 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 7 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected seroma (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaria (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mastitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coma scale abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adnexa uteri mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device breakage (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A, Neoadjuvant Phase: P+H IV (N=115) | Arm B, Neoadjuvant Phase: PH FDC SC (N=228) | Adjuvant Run-in Phase: PH FDC SC in Hospital (N=194) | Adjuvant Cross-Over Phase: PH FDC SC in Hospital (N=190) | Adjuvant Cross-Over Phase: PH FDC SC at Home (N=191) | Adjuvant Continuation Phase: PH FDC SC in Hospital (N=84) | Adjuvant Continuation Phase: PH FDC SC at Home (N=114) | Arm E, Adjuvant Phase: Trastuzumab Emtansine IV (N=117)
Anaemia (Blood and lymphatic system disorders) | 61 (82) | 96 (128) | 0 (0) | 5 (5) | 1 (1) | 1 (1) | 2 (2) | 20 (29)
Leukopenia (Blood and lymphatic system disorders) | 13 (29) | 26 (47) | 1 (1) | 1 (1) | 4 (4) | 3 (3) | 0 (0) | 13 (26)
Lymphopenia (Blood and lymphatic system disorders) | 8 (17) | 12 (18) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 8 (9)
Neutropenia (Blood and lymphatic system disorders) | 22 (36) | 60 (97) | 2 (2) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 22 (52)
Thrombocytopenia (Blood and lymphatic system disorders) | 12 (22) | 21 (33) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 25 (42)
Dry eye (Eye disorders) | 4 (4) | 15 (20) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (7) | 18 (21) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 6 (6)
Abdominal pain upper (Gastrointestinal disorders) | 9 (12) | 16 (20) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (9)
Constipation (Gastrointestinal disorders) | 14 (14) | 29 (45) | 2 (2) | 4 (4) | 5 (5) | 0 (0) | 1 (1) | 14 (15)
Diarrhoea (Gastrointestinal disorders) | 72 (145) | 147 (274) | 12 (14) | 9 (10) | 7 (8) | 3 (3) | 6 (6) | 7 (7)
Dyspepsia (Gastrointestinal disorders) | 14 (20) | 28 (32) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 (7) | 14 (15) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 64 (94) | 136 (245) | 5 (5) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 18 (26)
Stomatitis (Gastrointestinal disorders) | 13 (17) | 31 (37) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (7)
Vomiting (Gastrointestinal disorders) | 25 (34) | 57 (81) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 6 (8)
Asthenia (General disorders) | 18 (30) | 36 (54) | 3 (3) | 5 (5) | 3 (3) | 1 (1) | 0 (0) | 10 (11)
Fatigue (General disorders) | 41 (59) | 86 (131) | 9 (9) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 17 (18)
Influenza like illness (General disorders) | 3 (5) | 12 (12) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 4 (4)
Mucosal inflammation (General disorders) | 19 (26) | 35 (46) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Oedema peripheral (General disorders) | 9 (11) | 15 (17) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 3 (4)
Pain (General disorders) | 7 (8) | 11 (13) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 6 (6) | 27 (31) | 4 (4) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 2 (3)
COVID-19 (Infections and infestations) | 4 (4) | 10 (10) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 7 (7)
Upper respiratory tract infection (Infections and infestations) | 3 (5) | 15 (17) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 8 (8)
Urinary tract infection (Infections and infestations) | 13 (15) | 26 (31) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 9 (12)
Infusion related reaction (Injury, poisoning and procedural complications) | 14 (15) | 12 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 8 (8) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 27 (27) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 26 (26)
Alanine aminotransferase increased (Investigations) | 12 (16) | 26 (36) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 19 (24)
Aspartate aminotransferase increased (Investigations) | 11 (14) | 20 (27) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 26 (34)
Blood alkaline phosphatase increased (Investigations) | 5 (7) | 6 (6) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 10 (12)
Blood lactate dehydrogenase increased (Investigations) | 7 (10) | 8 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (11)
Neutrophil count decreased (Investigations) | 8 (17) | 30 (67) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 5 (9)
Platelet count decreased (Investigations) | 5 (8) | 10 (11) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 12 (14)
Weight decreased (Investigations) | 10 (11) | 17 (17) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 6 (6)
White blood cell count decreased (Investigations) | 4 (4) | 12 (21) | 4 (6) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 3 (7)
Decreased appetite (Metabolism and nutrition disorders) | 15 (15) | 45 (56) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 9 (9)
Dehydration (Metabolism and nutrition disorders) | 8 (9) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (16) | 23 (25) | 11 (11) | 5 (5) | 8 (10) | 0 (0) | 5 (5) | 31 (41)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 17 (18) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 6 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 13 (19) | 28 (35) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 3 (3) | 9 (16)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 10 (10) | 2 (2) | 3 (3) | 4 (4) | 3 (3) | 0 (0) | 6 (7)
Dizziness (Nervous system disorders) | 8 (8) | 11 (15) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 6 (6)
Dysgeusia (Nervous system disorders) | 13 (15) | 33 (36) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 16 (16) | 37 (44) | 9 (10) | 2 (2) | 3 (3) | 1 (1) | 6 (6) | 12 (13)
Neuropathy peripheral (Nervous system disorders) | 16 (16) | 41 (45) | 5 (5) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 14 (16)
Paraesthesia (Nervous system disorders) | 5 (6) | 21 (25) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 7 (9)
Peripheral sensory neuropathy (Nervous system disorders) | 9 (11) | 20 (20) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 17 (20)
Anxiety (Psychiatric disorders) | 8 (8) | 7 (7) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 5 (5)
Insomnia (Psychiatric disorders) | 11 (12) | 15 (15) | 4 (4) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 10 (10)
Dysuria (Renal and urinary disorders) | 4 (4) | 12 (13) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 21 (22) | 4 (4) | 2 (2) | 5 (5) | 1 (1) | 6 (6) | 9 (11)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 9 (10) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 (14) | 22 (31) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 14 (18)
Alopecia (Skin and subcutaneous tissue disorders) | 57 (60) | 124 (131) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (6) | 17 (18) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 6 (6) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 4 (5) | 13 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (10) | 15 (16) | 4 (4) | 4 (4) | 7 (8) | 3 (3) | 1 (1) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 11 (13) | 20 (21) | 2 (2) | 4 (4) | 1 (1) | 1 (1) | 1 (2) | 8 (8)
Flushing (Vascular disorders) | 6 (7) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 4 (4) | 14 (15) | 1 (1) | 5 (5) | 2 (2) | 0 (0) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2024-01-25): https://cdn.clinicaltrials.gov/large-docs/15/NCT05415215/Prot_000.pdf
  • Statistical Analysis Plan (2025-04-11): https://cdn.clinicaltrials.gov/large-docs/15/NCT05415215/SAP_001.pdf